CLINICAL TRIAL: NCT00611455
Title: A Double-blind, Randomized, Placebo Controlled, Parallel Group, Multi-center, Phase III Trial of Ofatumumab Investigating Clinical Efficacy in Adult Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Methotrexate Therapy
Brief Title: Investigating Clinical Efficacy of Ofatumumab in Adult Rheumatoid Arthritis (RA) Patients Who Had an Inadequate Response to MTX Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Ofatumumab IV trials in RA were prematurely terminated because GSK refocused clinical development of autoimmune indications on the subcutaneous delivery.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110635; GEN410 (Other: GENMAB)
Record Dates: First submitted 2008-01-16; First posted 2008-02-11 (Estimated); Results first posted 2011-10-28 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ofatumumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ofatumumab (Experimental): 1000 mL dilution of 35ml of ofatumumab in sterile, pyrogen free 0.9% NaCl. Each Treatment Cycle consisting of two 700mg IV infusions taken 14 days apart. A total of 8 infusions cycles given over a 144 week period
  Interventions: Drug: ofatumumab
- 1000 ml Saline (Placebo Comparator): 1000 mL dilution of 35ml of ofatumumab in sterile, pyrogen free 0.9% NaCl. Each Treatment Cycle consisting of two IV infusions taken 14 days apart. Only one placebo treatment cycle provided over a 24 week period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ofatumumab — 1000 mL dilution of 35ml of ofatumumab in sterile, pyrogen free 0.9% NaCl. Each Treatment Cycle consisting of two 700mg IV infusions taken 14 days apart. A total of 8 infusions cycles given over a 144 week period
  Arms: ofatumumab
Drug: Placebo — 1000 mL dilution of 35ml of ofatumumab in sterile, pyrogen free 0.9% NaCl. Each Treatment Cycle consisting of two IV infusions taken 14 days apart. Only one placebo treatment cycle provided over a 24 week period
  Arms: 1000 ml Saline

SUMMARY:
This is a phase III, double-blind, randomized, multicenter, and parallel group trial with a duration of 24 weeks, followed by a 120 week Open-label Period. the primary purpose of the study is to demonstrate the efficacy of ofatumumab in reducing clinical signs and symptoms in adult RA patients after a single course of ofatumumab.

DETAILED DESCRIPTION:
This study consists of a Double-blind , placebo controlled, and parallel group part with eligible patients enrolled into a 24 week Double-Blind Period, and randomized in a 1:1 ratio to receive ofatumumab (700mg x 2 infusions) or placebo ( saline x 2 infusions) in addition to their background methotrexate treatment. Patients who completed the 24 week Double-Blind period without receiving rescue DMARD treatment will be eligible to proceed into the 120 week Open-Label Period to receive repeat treatment courses with ofatumumab. In the Open-label Period ofatumumab treatment courses will be given at individualized time intervals only if a clinical response has been achieved following the previous treatment course, and followed by a subsequent worsening in disease activity . Patients who have completed the Open-Label Period or have withdrawn will enter a maximum 2 year Follow-up Period, or until their Bcells return to normal or to baseline levels, whichever occurs earlier.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years;
* Active disease at the time of screening as defined by:

  ≥ 8 swollen joints (of 66 joints assessed) and ≥ 8 tender joints (of 68 joints assessed), C-Reactive Protein (CRP) ≥ 1.0 mg/dL or Erythrocyte Sedimentation Rate (ESR) ≥ 22 mm/hour, DAS28≥3.2 (based on ESR);
* Inadequate response to previous or current methotrexate treatment;
* Treatment with methotrexate (MTX), 7.5-25 mg/week, for at least 12 weeks and at a stable dose for at least 4 weeks.

Exclusion Criteria

* Patients with a history of a rheumatic autoimmune disease other than RA or with significant systemic involvement secondary to RA;
* Previous exposure to biologic anti-rheumatic therapies, including investigational compounds;
* Previous exposure to biologic DMARDs; Chronic or ongoing active infectious disease requiring systemic treatment;
* Clinically significant cardiac disease; History of significant cerebrovascular disease;
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral psychiatric disease, or evidence of demyelinating disease;
* Known HIV positive; Serologic evidence of Hepatitis B infection; Positive test for Hepatitis C; Positive plasma / white cell JC Virus PCR;
* Serum IgG < lower limit of normal;
* Breast feeding women or women with a positive pregnancy test at screening;
* Current participation in any other interventional clinical study;
* Patients known or suspected of not being able to comply with a study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2008-01-01; Primary Completion 2009-06-08 (Actual); Study Completion 2013-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (41):
- Argentina (5):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Quilmes, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (5):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Maroochydore, Queensland
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Malvern, Victoria
  - GSK Investigational Site, Shenton Park, Western Australia
- Belgium (2):
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Merksem
- Chile (2):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- Czechia (3):
  - GSK Investigational Site, Ostrava Trebovice
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Zlín
- Hungary (2):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Győr
- Peru (2):
  - GSK Investigational Site, Callao
  - GSK Investigational Site, Lima
- Poland (4):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- GSK Investigational Site, Bucharest, Romania
- Russia (5):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- South Africa (2):
  - GSK Investigational Site, Gauteng
  - GSK Investigational Site, Parow
- Spain (4):
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
- United Kingdom (4):
  - GSK Investigational Site, Wigan, Lancashire
  - GSK Investigational Site, Cannock
  - GSK Investigational Site, Leytonstone, London
  - GSK Investigational Site, Maidstone

REFERENCES:
- [Background] Taylor PC, Quattrocchi E, Mallett S, Kurrasch R, Petersen J, Chang DJ. Ofatumumab, a fully human anti-CD20 monoclonal antibody, in biological-naive, rheumatoid arthritis patients with an inadequate response to methotrexate: a randomised, double-blind, placebo-controlled clinical trial. Ann Rheum Dis. 2011 Dec;70(12):2119-25. doi: 10.1136/ard.2011.151522. Epub 2011 Aug 22. PMID 21859685

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study OFA110635 was comprised of a 24-week Double-blind (DB) Period, followed by a 120-week Open-label (OL) Period. Participants who completed the OL Period, or who were withdrawn, entered a Follow-up (FU) period (approximately 2 years).
Groups:
- Placebo: Placebo was administered as two 1000 milliliter (ml) intravenous (IV) infusions, one at Day 0 and the other at Day 14, in addition to background methotrexate (MTX) treatment (7.5-25 milligrams [mg]/week [oral, intramuscular, or subcutaneous] for 24 weeks) in the DB Period.
- Ofatumumab 700 mg: Ofatumumab 700 mg (35 ml) was administered as two 1000 ml IV infusions, one at Day 0 and the other at Day 14, in addition to background MTX treatment (7.5 to 25 mg/week [oral, intramuscular, or subcutaneous] for 24 weeks) in the DB Period. Participants completing the 24-week DB Period without receiving rescue disease-modifying anti-rheumatic drug treatment were eligible to proceed into the 120-week OL Period to receive repeat ofatumumab treatment courses (at individualized time intervals if a clinical response had been achieved after the previous treatment course).
- Placebo or OFA 700 mg: FU Period: Participants randomized to DB treatment who completed the OL Period, who did not enter the OL Period, who did not qualify for retreatment, or who were withdrawn were to be followed until the number of B-cells and circulating IgG had returned to normal (according to the central laboratory) or Baseline levels or for a maximum of 2 years from the last scheduled visit in the DB or OL Periods, whichever occurred earlier. No investigational product was administered in the Follow-up Period.
Period: DB Treatment Period (24 Weeks)
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Started | 134 | 131 | 0
Completed | 121 | 117 | 0
Not Completed | 13 | 14 | 0
Not completed — Adverse Event | 2 | 8 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Protocol Violation | 4 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0
Not completed — Randomized in Error; Not Treated | 2 | 2 | 0
Not completed — Randomized, but Not Treated | 1 | 0 | 0
Period: OL Treatment Period (120 Weeks)
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Started | 0 | 231 (118 participants received OFA during the DB Period; 113 received placebo during the DB Period.) | 0
Completed | 0 | 52 | 0
Not Completed | 0 | 179 | 0
Not completed — Adverse Event | 0 | 17 | 0
Not completed — Lack of Efficacy | 0 | 9 | 0
Not completed — Protocol Violation | 0 | 3 | 0
Not completed — Protocol-defined Stopping Criteria Met | 0 | 12 | 0
Not completed — Study Closed/Terminated | 0 | 110 | 0
Not completed — Lost to Follow-up | 0 | 5 | 0
Not completed — Physician Decision | 0 | 5 | 0
Not completed — Withdrawal by Subject | 0 | 18 | 0
Period: Follow-up Period (Approximately 2 Years)
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Started | 0 | 0 | 260 (These participants received at least one infusion of placebo or ofatumumab.)
Completed | 0 | 0 | 49
Not Completed | 0 | 0 | 211
Not completed — Adverse Event | 0 | 0 | 30
Not completed — Lack of Efficacy | 0 | 0 | 12
Not completed — Protocol Violation | 0 | 0 | 4
Not completed — Protocol-defined Stopping Criteria Met | 0 | 0 | 23
Not completed — Study Closed/Terminated | 0 | 0 | 80
Not completed — Lost to Follow-up | 0 | 0 | 13
Not completed — Withdrawal by Subject | 0 | 0 | 49

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo was administered as two 1000 milliliter (ml) intravenous (IV) infusions, one at Day 0 and the other at Day 14, in addition to background methotrexate (MTX) treatment (7.5 to 25 milligrams [mg]/week [oral, intramuscular, or subcutaneous] for 24 weeks).
- Ofatumumab 700 mg: Ofatumumab 700 mg (35 ml) was administered as two 1000 ml IV infusions, one at Day 0 and the other at Day 14, in addition to background MTX treatment (7.5 to 25 mg/week [oral, intramuscular, or subcutaneous] for 24 weeks).
- Total: Total of all reporting groups
Arm/Group | Placebo | Ofatumumab 700 mg | Total
Number analyzed (Participants) | 131 | 129 | 260
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics are reported for members of the Intent-to-Treat (ITT) Population, comprised of all randomized participants who were exposed to investigational product irrespective of their compliance to the planned course of treatment. Participants were analyzed according to their randomized treatment.
  Years | 53.6 (11.50) | 51.7 (11.24) | 52.7 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics are reported for members of the ITT Population, comprised of all randomized participants who were exposed to investigational product irrespective of their compliance to the planned course of treatment. Participants were analyzed according to their randomized treatment.
  Participants
    Female | 108 | 106 | 214
    Male | 23 | 23 | 46
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics are reported for members of the ITT Population, comprised of all randomized participants who were exposed to investigational product irrespective of their compliance to the planned course of treatment. Participants were analyzed according to their randomized treatment.
  participants
    Hispanic/Latino | 52 | 51 | 103
    Not Hispanic/Latino | 79 | 78 | 157

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 20% Improvement From Baseline in Their American College of Rheumatology (ACR) Score (ACR20) at Week 24
Description: The ACR score was based on improvement from baseline in tender (TJC) and swollen joint counts (SJC). A participant had achieved ACR20 if he experienced >=20% improvement from baseline in TJC and SJC and a >=20% improvement from baseline in 3 out of 5 of the following assessments: participant pain assessment on a 100 millimeter (mm) visual analog scale (VAS), participant global assessment on a 100 mm VAS scale, physician global assessment on a 100 mm VAS scale, participant self-assessed disability, and C-reactive protein.
Time Frame: Baseline and Week 24
Population: Intent-to-Treat (ITT) Population: all randomized participants who were exposed to investigational product irrespective of their compliance to the planned course of treatment. Participants were analyzed according to their randomized treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 131 | 129
participants | 35 | 64
Statistical Analysis 1: Comparison: Placebo vs Ofatumumab 700 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.86, 95% CI 2-sided [1.67 to 4.91]

2. Secondary Outcome: Number of Participants With a 20% Improvement From Baseline in Their American College of Rheumatology (ACR) Score (ACR20) at Weeks 4, 8, 12, 16, and 20
Description: as for outcome 1
Time Frame: Baseline and Weeks 4, 8, 12, 16, and 20
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 131 | 129
participants
  Week 4 | 42 | 52
  Week 8 | 43 | 66
  Week 12 | 44 | 71
  Week 16 | 38 | 67
  Week 20 | 40 | 62

3. Secondary Outcome: Number of Participants With a 50% Improvement From Baseline in Their ACR Score (ACR50) at Weeks 4, 8, 12, 16, 20, and 24
Description: The ACR score was based on improvement from baseline in tender (TJC) and swollen joint counts (SJC). A participant had achieved ACR50 if he experienced >=50% improvement from baseline in TJC and SJC and a >=50% improvement from baseline in 3 out of 5 of the following assessments: participant pain assessment on a 100 millimeter (mm) visual analog scale (VAS), participant global assessment on a 100 mm VAS scale, physician global assessment on a 100 mm VAS scale, participant self-assessed disability, and C-reactive protein.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 131 | 129
participants
  Week 4 | 13 | 14
  Week 8 | 12 | 23
  Week 12 | 14 | 36
  Week 16 | 13 | 37
  Week 20 | 19 | 31
  Week 24 | 14 | 35

4. Secondary Outcome: Number of Participants With a 70% Improvement From Baseline in Their ACR Score (ACR70) at Weeks 4, 8, 12, 16, 20, and 24
Description: The ACR score was based on improvement from baseline in tender (TJC) and swollen joint counts (SJC). A participant had achieved ACR70 if he experienced >=70% improvement from baseline in TJC and SJC and a >=70% improvement from baseline in 3 out of 5 of the following assessments: participant pain assessment on a 100 millimeter (mm) visual analog scale (VAS), participant global assessment on a 100 mm VAS scale, physician global assessment on a 100 mm VAS scale, participant self-assessed disability, and C-reactive protein.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 131 | 129
participants
  Week 4 | 6 | 4
  Week 8 | 3 | 10
  Week 12 | 6 | 19
  Week 16 | 5 | 18
  Week 20 | 6 | 18
  Week 24 | 3 | 17

5. Secondary Outcome: Median ACRn at Weeks 4, 8, 12, 16, 20, and 24
Description: ACRn = the largest integer n for which a participant (par.) met the criteria requiring an improvement of n%. ACRn is a measure characterizing percent (%) improvement from baseline (IFBL). A par. with an ACRn of X had an improvement of >=X% in tender/swollen joints (TJC/SJC), and an improvement of >=X% in 3 of the 5 parameters (patient [pt] pain assessment, pt global assessment [GA], physician GA, pt self-assessed disability, acute phase reactant). ACRn = minimum(TJC % IFBL, SJC % IFBL, composite measure % IFBL). Composite measure % IFBL is the 3rd highest value of % IFBL for the 5 parameters.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population. Missing data were imputed using last observation carried forward (LOCF). Analysis included those participants in the ITT Population with at least one post-baseline efficacy assessment.
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 130 | 126
percent change
  Week 4, n=129, 124 | 6.0 [-77 to 85] | 13.0 [-98 to 92]
  Week 8, n=130, 126 | 5.5 [-250 to 86] | 22.0 [-264 to 84]
  Week 12, n=130, 126 | 0.5 [-200 to 85] | 25.0 [-73 to 100]
  Week 16, n=130, 126 | 0.0 [-210 to 85] | 26.0 [-138 to 93]
  Week 20, n=130, 126 | 4.0 [-185 to 90] | 21.0 [-74 to 92]
  Week 24, n=130, 126 | -2.5 [-272 to 90] | 21.0 [-87 to 95]

6. Secondary Outcome: Mean Disease Activity Score Based on 28 Joints (DAS28) at Weeks 4, 8, 12, 16, 20, and 24 Using C-reactive Protein (CRP) as the Acute Phase Reactant (APR)
Description: The DAS28 is a clinical index of rheumatoid arthritis disease activity (DA) that combines information from swollen and tender joints (jts.), the APR, and general health (patient global assessment). The following jts. were assessed on both sides of the body: shoulder, elbow, wrist, metacarpophalangeal (5 per side), proximal interphalangeal (5 per side), and knee. The level of DA can be interpreted as low (DAS28<=3.2), moderate (3.2<DAS28<=5.1), or high (DAS28>5.1); total score, 0-9.4. A DAS28 <2.6 corresponds to remission. APRs are a class of proteins that are useful markers for inflammation.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population. Missing data were imputed using LOCF. Analysis included those participants in the ITT Population with at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 130 | 126
scores on a scale
  Week 4, n=129, 124 | 4.78 (1.241) | 4.74 (1.099)
  Week 8, n=130, 126 | 4.75 (1.205) | 4.41 (1.285)
  Week 12, n=130, 126 | 4.66 (1.333) | 4.14 (1.367)
  Week 16, n=130, 126 | 4.78 (1.327) | 4.11 (1.296)
  Week 20, n=130, 126 | 4.78 (1.387) | 4.13 (1.395)
  Week 24, n=130, 126 | 4.98 (1.437) | 4.12 (1.270)

7. Secondary Outcome: Change From Baseline in DAS28 at Weeks 4, 8, 12, 16, 20, and 24 Using CRP as the Acute Phase Reactant
Description: The DAS28 is a clinical index of RA disease activity that combines information from swollen joints, tender joints, the acute phase reactant, and general health (patient global assessment). Change from baseline in DAS28 is calculated as the Week 4, 8, 12, 16, 20, and 24 values minus the baseline value.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 130 | 126
scores on a scale
  Week 4, n=129, 124 | -0.84 (1.053) | -1.09 (0.886)
  Week 8, n=130, 126 | -0.88 (0.992) | -1.41 (1.112)
  Week 12, n=130, 126 | -0.97 (1.221) | -1.69 (1.255)
  Week 16, n=130, 126 | -0.85 (1.194) | -1.72 (1.166)
  Week 20, n=130, 126 | -0.85 (1.215) | -1.70 (1.262)
  Week 24, n=130, 126 | -0.65 (1.218) | -1.71 (1.201)

8. Secondary Outcome: Mean DAS28 at Weeks 4, 8, 12, 16, 20, and 24 Using Erythrocyte Sedimentation Rate (ESR) as the Acute Phase Reactant
Description: as for outcome 6
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 130 | 126
scores on a scale
  Week 4, n=129, 124 | 5.48 (1.332) | 5.51 (1.127)
  Week 8, n=130, 126 | 5.43 (1.289) | 5.14 (1.276)
  Week 12, n=130, 126 | 5.31 (1.349) | 4.83 (1.358)
  Week 16, n=130, 126 | 5.43 (1.329) | 4.81 (1.310)
  Week 20, n=130, 126 | 5.41 (1.414) | 4.77 (1.427)
  Week 24, n=130, 126 | 5.67 (1.439) | 4.84 (1.360)

9. Secondary Outcome: Change From Baseline in DAS28 at Weeks 4, 8, 12, 16, 20, and 24 Using ESR as the Acute Phase Reactant
Description: as for outcome 7
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 130 | 126
scores on a scale
  Week 4, n=129, 124 | -0.92 (1.106) | -1.08 (0.891)
  Week 8, n=130, 126 | -0.97 (1.048) | -1.46 (1.092)
  Week 12, n=130, 126 | -1.10 (1.211) | -1.77 (1.257)
  Week 16, n=130, 126 | -0.97 (1.183) | -1.79 (1.189)
  Week 20, n=130, 126 | -0.99 (1.175) | -1.83 (1.304)
  Week 24, n=130, 126 | -0.73 (1.203) | -1.76 (1.264)

10. Secondary Outcome: Number of Participants With the Indicated European League Against Rheumatism (EULAR) Response at Weeks 4, 8, 12, 16, 20, and 24 Using CRP as the Acute Phase Reactant
Description: The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 <=3.2; moderate responders: change from baseline >1.2 with DAS28 <=3.2 to >5.1 or change from baseline >0.6 to <=1.2 with DAS28 <=3.2 to <=5.1); non-responders: change from baseline <=0.6 or change from baseline >0.6 and <=1.2 with DAS28 >5.1.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 130 | 126
participants
  Week 4, Good; n=129, 124 | 15 | 12
  Week 4, Moderate; n=129, 124 | 41 | 63
  Week 4, None; n=129, 124 | 73 | 49
  Week 8, Good; n=130, 126 | 16 | 22
  Week 8, Moderate; n=130, 126 | 49 | 62
  Week 8, None; n=130, 126 | 65 | 42
  Week 12, Good; n=130, 126 | 17 | 32
  Week 12, Moderate; n=130, 126 | 51 | 56
  Week 12, None; n=130, 126 | 62 | 38
  Week 16, Good; n=130, 126 | 16 | 32
  Week 16, Moderate; n=130, 126 | 51 | 58
  Week 16, None; n=130, 126 | 63 | 36
  Week 20, Good; n=130, 126 | 17 | 34
  Week 20, Moderate; n=130, 126 | 41 | 52
  Week 20, None; n=130, 126 | 72 | 40
  Week 24, Good; n=130, 126 | 18 | 32
  Week 24, Moderate; n=130, 126 | 37 | 60
  Week 24, None; n=130, 126 | 75 | 34

11. Secondary Outcome: Number of Participants With the Indicated European League Against Rheumatism (EULAR) Response at Weeks 4, 8, 12, 16, 20, and 24 Using ESR as the Acute Phase Reactant
Description: as for outcome 10
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 130 | 126
participants
  Week 4, Good; n=129, 124 | 6 | 5
  Week 4, Moderate; n=129, 124 | 49 | 50
  Week 4, None; n=129, 124 | 74 | 69
  Week 8, Good; n=130, 126 | 7 | 8
  Week 8, Moderate; n=130, 126 | 53 | 67
  Week 8, None; n=130, 126 | 70 | 51
  Week 12, Good; n=130, 126 | 7 | 17
  Week 12, Moderate; n=130, 126 | 57 | 63
  Week 12, None; n=130, 126 | 66 | 46
  Week 16, Good; n=130, 126 | 4 | 15
  Week 16, Moderate; n=130, 126 | 58 | 70
  Week 16, None; n=130, 126 | 68 | 41
  Week 20, Good; n=130, 126 | 8 | 22
  Week 20, Moderate; n=130, 126 | 45 | 63
  Week 20, None; n=130, 126 | 77 | 41
  Week 24, Good; n=130, 126 | 4 | 14
  Week 24, Moderate; n=130, 126 | 44 | 67
  Week 24, None; n=130, 126 | 82 | 45

12. Secondary Outcome: Number of Participants Classified as Responders at Week 24 According to the Self-Assessed Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The HAQ-DI is a 20-question instrument used to assess the degree of difficulty a participant had in accomplishing tasks in 8 functional areas (FAs): dressing, arising, eating, walking, hygiene, reaching, gripping, and errands/chores. Responses for each FA were scored from 0 (no difficulty) to 3 (inability to perform a task). The total score (range of 0-3) was calculated by adding the 8 individual FA scores, then dividing this sum by the total number of components answered. Responders were defined as participants achieving an improvement from baseline in the HAQ-DI score at Week 24 of >=0.22.
Time Frame: Week 24
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 117 | 112
participants | 59 | 74

13. Secondary Outcome: Number of Participants With Clinical Remission at Week 24
Description: Participants achieving clinical remission were defined as those with a low disease activity, i.e., DAS28 score (using CRP) <2.6 at Week 24.
Time Frame: Week 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 131 | 129
participants | 7 | 13

14. Secondary Outcome: Change From Baseline in Tender Joint Count at Week 24
Description: Change from baseline in tender joint count was calculated as the Week 24 count minus the baseline count. A total of 68 joints were assessed. Joints were classified as either tender or not tender by an independent assessor, who had documented experience in performing joint assessments.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Median (Full Range); unit: number of tender joints
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 130 | 126
number of tender joints | -5 [-38 to 36] | -12 [-52 to 20]

15. Secondary Outcome: Change From Baseline in Swollen Joint Count at Week 24
Description: Change from baseline in swollen joint count was calculated as the Week 24 count minus the baseline count. A total of 66 joints were assessed. Joints were classified as either swollen or not swollen by an independent assessor, who had documented experience in performing joint assessments.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Median (Full Range); unit: number of swollen joints
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 130 | 126
number of swollen joints | -4.50 [-24 to 16] | -8.00 [-43 to 12]

16. Secondary Outcome: Change From Baseline in the Participant-assessed Pain Score at Week 24
Description: A horizontal VAS of 100 mm was used to report the participant's level of joint pain. The scale ranged from 0 (no pain) to 100 (unbearable pain). Participants were instructed to draw a vertical line through the horizontal line to indicate how much joint pain they had. The distance from the "no pain" end to the vertical line drawn by the participant was the joint pain score. Change from baseline was calculated as the Week 24 value minus the baseline value.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 128 | 119
scores on a scale | -5 [-93 to 54] | -22 [-95 to 35]

17. Secondary Outcome: Change From Baseline in Participant-assessed Global Disease Score at Week 24
Description: The participant used a horizontal VAS of 100 mm for overall assessment of disease. The scale ranged from 0 (very well) to 100 (very poor). Participants were instructed to draw a vertical line through the horizontal line to indicate the state of the arthritis. The distance from the "very well" end to the vertical line drawn by the participant was the global disease assessment score. Change from baseline in participant-assessed global disease was calculated as the Week 24 value minus the baseline value.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 130 | 126
scores on a scale | -6.0 [-76 to 57] | -16.5 [-83 to 28]

18. Secondary Outcome: Change From Baseline in the Physician-assessed Global Disease Score at Week 24
Description: The physician used a horizontal VAS of 100 mm for overall assessment of disease. The scale ranged from 0 (very well) to 100 (very poor). Physicians were instructed to draw a vertical line through the horizontal line to indicate the state of the arthritis. The distance from the "very well" end to the vertical line drawn by the participant was the global disease assessment score. Change from baseline in the physician-assessed global disease was calculated as the Week 24 value minus the baseline value.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 130 | 124
scores on a scale | -9.50 [-70 to 37] | -20.50 [-77 to 17]

19. Secondary Outcome: Change From Baseline in HAQ-DI Score at Week 24
Description: The self-assessed HAQ-DI is a 20-question instrument used to assess the degree of difficulty a participant had in accomplishing tasks in 8 functional areas (FAs): dressing, arising, eating, walking, hygiene, reaching, gripping, and errands/chores. Responses for each FA were scored from 0 (no difficulty) to 3 (inability to perform a task). The total score (range of 0-3) was calculated by adding the 8 individual FA scores, then dividing this sum by the total number of components answered. Change from baseline was calculated as the value at Week 24 minus the baseline value.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 123 | 122
scores on a scale | -0.25 [-2.4 to 1.3] | -0.38 [-2.4 to 1.0]

20. Secondary Outcome: Change From Baseline in CRP at Week 24
Description: Blood samples for the determination of CRP were taken at pre-specified visits and were sent to the central laboratory for analysis. Change from Baseline in CRP was calculated as the Week 24 value minus the baseline value. CRP is an acute-phase protein whose plasma concentration increases in response to inflammation. CRP is a useful marker of inflammation.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Median (Full Range); unit: milligrams per liter (mg/L)
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 130 | 126
milligrams per liter (mg/L) | -0.10 [-55.1 to 96.2] | -4.85 [-96.2 to 30.2]

21. Secondary Outcome: Change From Baseline in ESR at Week 24
Description: ESR is measured by a blood test that shows the rate at which red blood cells sediment in a period of 1 hour. Blood samples for the determination of ESR were taken at pre-specified visits and were measured immediately at the trial site. Change from baseline in ESR was calculated as the Week 24 value minus the baseline value.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Median (Full Range); unit: millimeters per hour (mm/hr)
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 130 | 126
millimeters per hour (mm/hr) | -5 [-57 to 89] | -15 [-85 to 34]

22. Secondary Outcome: Change From Baseline in the Short-Form 36 (SF-36v2) Norm-based Scores for Physical Component Summary and Physical Items at Week 24
Description: The SF-36v2 is a standardized questionnaire used to measure overall subjective health status by measuring 8 health-related parameters (each scored from 0 [poorer health] to 100 [better health]): body pain, general mental health (MH), perception of general health, physical functioning, role limitations (RL) caused by mental condition, RL caused by a physical condition, social functioning, and vitality. It yields an 8-scale profile of functional health and well-being scores, as well as psychometrically based physical and MH summary measures and a preference-based health utility index.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 117 | 116
scores on a scale
  Physical Component Summary | 4.21 (1.048) | 6.69 (1.031)
  Physical Functioning | 3.14 (1.125) | 5.70 (1.100)
  Role Physical | 5.43 (1.259) | 6.64 (1.231)
  Bodily Pain | 3.63 (1.197) | 8.28 (1.170)
  General Health | 2.28 (1.033) | 4.08 (1.011)

23. Secondary Outcome: Change From Baseline in the SF-36v2 Norm-based Scores for Mental Component Summary and Mental Items at Week 24
Description: as for outcome 22
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 117 | 116
scores on a scale
  Mental Component Summary | 1.57 (1.308) | 4.60 (1.272)
  Vitality | 2.46 (1.169) | 7.26 (1.154)
  Social Functioning | 3.56 (1.361) | 4.98 (1.331)
  Role Emotional | 2.23 (1.612) | 4.93 (1.563)
  Mental Health | 2.92 (1.278) | 5.40 (1.249)

24. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy (FACIT) Questionnaire Score at Week 24
Description: The FACIT-F score has a valid range of values from 0 to 52, with a higher score indicating a lower burden of fatigue. The subset determining fatigue contains 13 questions. Responses to each question were scored from 0, indicating "Not at all fatigued," to 4, indicating "Very much fatigued."
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 111 | 114
scores on a scale | 2 [-37 to 27] | 6 [-19 to 42]

25. Secondary Outcome: Change From Baseline in Levels of Anti-CCP, RF-IgA, RF-IgG, and RF-IgM at Week 24
Description: The following biomarkers were assessed: Anti-Cyclic Citrullinated Peptide 3 antibody (Anti-CCP), Rheumatoid factor IgA (RF-IgA), RF IgG (RF-IgG), and RF IgM (RF-IgM). Measurements of RF were used to characterize participants' disease activity and immune status. Anti-CCP was used to characterize the disease type and the immune status of the participants. Assessments for which results were below the lower limit of quantification (LLQ) were reported using a value of LLQ/2. Assessments for which results were above the upper limit of quantification (ULQ) were reported using a value of ULQ.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Median (Full Range); unit: Units/Liter
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 120 | 115
Units/Liter
  Anti-CCP, n=120, 115 | 0.0 [-1613 to 4042] | -138.0 [-13000 to 762]
  RF-IgA, n=119, 110 | 0.0 [-79 to 72] | -3 [-93 to 3]
  RF-IgG, n=119, 110 | 0.0 [-71 to 58] | -4.8 [-87 to 9]
  RF-IgM, n=119, 110 | 0.0 [-68 to 98] | -6.3 [-93 to 98]

26. Secondary Outcome: Change From Baseline in Levels of IL-6 and Serum Amyloid A at Week 24
Description: The following biomarkers were assessed: Interleukin 6 (IL-6) and Serum Amyloid A. These biomarkers were used to further characterize disease activity.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Median (Full Range); unit: nanogram per liter (ng/l)
Arm/Group | Placebo | Ofatumumab 700 mg
Number analyzed (Participants) | 120 | 115
nanogram per liter (ng/l)
  IL-6, n=119, 115 | -0.410 [-131.26 to 2632.66] | -4.040 [-106.98 to 63.44]
  Serum Amyloid A, n=120, 114 | -10850.5 [-1680680 to 3374580] | -53513.5 [-3724434 to 931790]

27. Secondary Outcome: Minimum DAS28-ESR Score During the Double-blind (DB) and Open-label (OL) Periods, by Ofatumumab Treatment Course
Description: The DAS28 is a clinical index of rheumatoid arthritis disease activity that combines information from swollen and tender joints (jts.), the APR, and general health (patient global assessment). The following jts. were assessed on both sides of the body: shoulder, elbow, wrist, metacarpophalangeal (5 per side), proximal interphalangeal (5 per side), and knee. The level of disease activity can be interpreted as low (DAS28<=3.2), moderate (3.2<DAS28<=5.1), or high (DAS28>5.1); total score, 0-9.4. A DAS28 <2.6 corresponds to remission. The values summarized are the minimum DAS28 score (i.e. lowest level of disease activity) achieved by each participant within the first 24 weeks of each treatment course (TC), assessed using erythrocyte sedimentation rate (ESR; rate at which red blood cells sediment in 1 hour).
Time Frame: First 24 weeks of each treatment course (assessed up to Week 144)
Population: As Treated (AT) Population: all participants who received at least one infusion of ofatumumab in the DB and/or OL Period. Only those participants contributing values at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 243 | 0
Scores on a scale
  TC 1, n=0, 243, 0 |  | 4.01 (1.396) |
  TC 2, n=0, 198, 0 |  | 3.59 (1.227) |
  TC 3, n=0, 136, 0 |  | 3.36 (1.225) |
  TC 4, n=0, 72, 0 |  | 3.50 (1.175) |
  TC 5, n=0, 31, 0 |  | 3.34 (1.326) |
  TC 6, n=0, 11, 0 |  | 3.82 (1.588) |
  TC 7, n=0, 2, 0 |  | 5.34 (1.038) |

28. Secondary Outcome: Minimum DAS28-CRP Score During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The DAS28 is a clinical index of rheumatoid arthritis disease activity that combines information from swollen and tender joints (jts.), the APR, and general health (patient global assessment). The following jts. were assessed on both sides of the body: shoulder, elbow, wrist, metacarpophalangeal (5 per side), proximal interphalangeal (5 per side), and knee. The level of disease activity can be interpreted as low (DAS28<=3.2), moderate (3.2<DAS28<=5.1), or high (DAS28>5.1); total score, 0-9.4. A DAS28 <2.6 corresponds to remission. The values summarized are the minimum DAS28 score (i.e. lowest level of disease activity) achieved by each participant within the first 24 weeks of each treatment course, assessed using C-reactive Protein (CRP: used to monitor acute inflammatory phases of rheumatoid arthritis).
Time Frame: First 24 weeks of each treatment course (assessed up to Week 144)
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 243 | 0
scores on a scale
  TC 1, n=0, 243, 0 |  | 3.43 (1.321) |
  TC 2, n=0, 198, 0 |  | 3.09 (1.142) |
  TC 3, n=0, 136, 0 |  | 2.86 (1.156) |
  TC 4, n=0, 72, 0 |  | 2.94 (1.161) |
  TC 5, n=0, 31, 0 |  | 2.90 (1.362) |
  TC 6, n=0, 11, 0 |  | 3.39 (1.401) |
  TC 7, n=0, 2, 0 |  | 4.55 (1.003) |

29. Secondary Outcome: Minimum Change From Baseline in the DAS28-ESR Score, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The level of rheumatoid arthritis disease activity based on the DAS28 score is defined as low if DAS28 <=3.2, moderate if 3.2< DAS28 <=5.1, or high if DAS28 > 5.1. A DAS28 <2.6 corresponds to clinical remission. The values summarized are the minimum change from baseline DAS28 score (i.e. greatest change in disease activity during the treatment course) achieved by each participant within the first 24 weeks of each treatment course, assessed by using ESR. Baseline score was determined at the start of each treatment course. For change from baseline, participants had to have both a baseline DAS28 value for the treatment course (i.e., the latest value on or before the date of infusion A of the treatment course, providing it was done within a 14 day window prior to the date of infusion A) and a DAS28 value during the treatment course (i.e., during first 24 weeks of each treatment course). Change from baseline was calculated as the value during the treatment course minus the baseline value.
Time Frame: First 24 weeks of each treatment course (assessed up to Week 144)
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 238 | 0
scores on a scale
  TC 1, n=0, 238, 0 |  | -2.32 (1.192) |
  TC 2, n=0, 194, 0 |  | -1.77 (1.072) |
  TC 3, n=0, 129, 0 |  | -1.77 (1.203) |
  TC 4, n=0, 69, 0 |  | -1.47 (1.065) |
  TC 5, n=0, 31, 0 |  | -1.77 (1.015) |
  TC 6, n=0, 11, 0 |  | -1.45 (0.845) |
  TC 7, n=0, 2, 0 |  | -0.07 (0.696) |

30. Secondary Outcome: Minimum Change From Baseline in the DAS28-CRP Score, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The level of rheumatoid arthritis disease activity based on the DAS28 score is defined as low if DAS28 <=3.2, moderate if 3.2< DAS28 <=5.1, or high if DAS28 > 5.1. A DAS28 <2.6 corresponds to clinical remission. The values summarized are the minimum change from baseline DAS28 score (i.e. greatest change in disease activity during the treatment course) achieved by each participant within the first 24 weeks of each treatment course, assessed by using CRP. Baseline score was determined at the start of each treatment course. For change from baseline, participants had to have both a baseline DAS28 value for the treatment course (i.e., the latest value on or before the date of infusion A of the treatment course, providing it was done within a 14 day window prior to the date of infusion A) and a DAS28 value during the treatment course (i.e., during first 24 weeks of each treatment course). Change from baseline was calculated as the value during the treatment course minus the baseline value.
Time Frame: First 24 weeks of each treatment course (assessed up to Week 144)
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 237 | 0
scores on a scale
  TC 1, n=0, 237, 0 |  | -2.15 (1.166) |
  TC 2, n=0, 193, 0 |  | -1.55 (1.020) |
  TC 3, n=0, 125, 0 |  | -1.67 (1.144) |
  TC 4, n=0, 69, 0 |  | -1.40 (1.081) |
  TC 5, n=0, 31, 0 |  | -1.61 (1.036) |
  TC 6, n=0, 11, 0 |  | -1.33 (0.710) |
  TC 7, n=0, 2, 0 |  | -0.05 (0.200) |

31. Secondary Outcome: Number of Participants Who Achieved Remission or Low Disease Activity Based on DAS28 (Using ESR), During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The DAS28 is a clinical index of rheumatoid arthritis disease activity that combines information from swollen and tender joints (jts.), the APR, and general health (patient global assessment). The following jts. were assessed on both sides of the body: shoulder, elbow, wrist, metacarpophalangeal (5 per side), proximal interphalangeal (5 per side), and knee. The level of disease activity can be interpreted as low (DAS28<=3.2), moderate (3.2<DAS28<=5.1), or high (DAS28>5.1); total score, 0-9.4. A DAS28 <2.6 corresponds to remission. Remission is defined as a DAS28 score <2.6 at any time during the first 24 weeks of each treatment course. Low disease activity is defined as a DAS28 score >=2.6 and <3.2 at any time during the first 24 weeks of each treatment course.
Time Frame: First 24 weeks of each treatment course (assessed up to Week 144)
Population: AT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 243 | 0
participants
  TC 1, Remission, n=0, 243, 0 |  | 38 |
  TC 1, Low Disease Activity, n=0, 243, 0 |  | 33 |
  TC 2, Remission, n=0, 198, 0 |  | 47 |
  TC 2, Low Disease Activity, n=0, 198, 0 |  | 33 |
  TC 3, Remission, n=0, 136, 0 |  | 40 |
  TC 3, Low Disease Activity, n=0, 136, 0 |  | 31 |
  TC 4, Remission, n=0, 72, 0 |  | 15 |
  TC 4, Low Disease Activity, n=0, 72, 0 |  | 20 |
  TC 5, Remission, n=0, 31, 0 |  | 13 |
  TC 5, Low Disease Activity, n=0, 31, 0 |  | 4 |
  TC 6, Remission, n=0, 11, 0 |  | 3 |
  TC 6, Low Disease Activity, n=0, 11, 0 |  | 1 |
  TC 7, Remission, n=0, 2, 0 |  | 0 |
  TC 7, Low Disease Activity, n=0, 2, 0 |  | 0 |

32. Secondary Outcome: Number of Participants Who Achieved Remission or Low Disease Activity Based on DAS28 (Using CRP), During the DB and OL Periods, by Ofatumumab Treatment Course
Description: as for outcome 31
Time Frame: First 24 weeks of each treatment course (assessed up to Week 144)
Population: AT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 243 | 0
participants
  TC 1, Remission, n=0, 243, 0 |  | 71 |
  TC 1, Low Disease Activity, n=0, 243, 0 |  | 44 |
  TC 2, Remission, n=0, 198, 0 |  | 71 |
  TC 2, Low Disease Activity, n=0, 198, 0 |  | 36 |
  TC 3, Remission, n=0, 136, 0 |  | 63 |
  TC 3, Low Disease Activity, n=0, 136, 0 |  | 21 |
  TC 4, Remission, n=0, 72, 0 |  | 30 |
  TC 4, Low Disease Activity, n=0, 72, 0 |  | 11 |
  TC 5, Remission,n=0, 31, 0 |  | 14 |
  TC 5, Low Disease Activity,n=0, 31, 0 |  | 4 |
  TC 6, Remission,n=0, 11, 0 |  | 4 |
  TC 6, Low Disease Activity,n=0, 11, 0 |  | 2 |
  TC 7, Remission, n=0, 2, 0 |  | 0 |
  TC 7, Low Disease Activity, n=0, 2, 0 |  | 0 |

33. Secondary Outcome: Time to Retreatment, by Ofatumumab Treatment Course
Description: Time to retreatment is defined as the time in days between infusion A of each treatment course and infusion A of the following treatment course. For participants randomized to ofatumumab in the Double-blind Period, Treatment Course 1 refers to the course of ofatumumab received in the Double-blind Period. The minimum period allowed per protocol before retreatment was 24 weeks (end of Double-blind Period). For participants randomized to placebo in the Double-blind Period, Treatment Course 1 refers to the first course of ofatumumab received in the Open-label Period. The minimum period allowed per protocol before retreatment during the Open-label Period was 16 weeks.
Time Frame: From Baseline up to Week 144
Population: AT Population. Only those participants who were retreated from Week 24 were analyzed.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 198 | 0
Weeks
  TC 1, n=0, 198, 0 |  | 34.26 (15.828) |
  TC 2, n=0, 136, 0 |  | 34.50 (15.151) |
  TC 3, n=0, 72, 0 |  | 28.83 (10.713) |
  TC 4, n=0, 31, 0 |  | 20.82 (6.952) |
  TC 5, n=0, 11, 0 |  | 19.94 (5.411) |
  TC 6, n=0, 2, 0 |  | 17.86 (0.404) |
  TC 7, n=0, 0, 0 |  | NA (NA) — Data are not available because there was no subsequent treatment course after Treatment Course 7. |

34. Secondary Outcome: Number of Participants With Any On-treatment Adverse Event or Serious Adverse Event, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; or is a congenital anomaly/birth defect. Medical or scientific judgment should have been exercised in other situations. Refer to the general AE/SAE module for a list of AEs (occurring at a frequency threshold >=2%) and SAEs.
Time Frame: First treatment (Day 0) until the participant terminated the trial, assessed up to Week 144
Population: AT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 243 | 0
Participants
  Any AE, TC 1, n=0, 243, 0 |  | 212 |
  Any AE, TC 2, n=0, 198, 0 |  | 151 |
  Any AE, TC 3, n=0, 136, 0 |  | 91 |
  Any AE, TC 4, n=0, 72, 0 |  | 43 |
  Any AE, TC 5, n=0, 31, 0 |  | 14 |
  Any AE, TC 6, n=0, 11, 0 |  | 5 |
  Any AE, TC 7, n=0, 2, 0 |  | 0 |
  Any SAE, TC 1, n=0, 243, 0 |  | 14 |
  Any SAE, TC 2, n=0, 198, 0 |  | 19 |
  Any SAE, TC 3, n=0, 136, 0 |  | 12 |
  Any SAE, TC 4, n=0, 72, 0 |  | 4 |
  Any SAE, TC 5, n=0, 31, 0 |  | 1 |
  Any SAE, TC 6, n=0, 11, 0 |  | 0 |
  Any SAE, TC 7, n=0, 2, 0 |  | 0 |

35. Secondary Outcome: Number of Participants With a CD19+ Cell Count Greater Than or Equal to the Lower Limit of Normal or the Baseline Value at the Indicated Time Point, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The number of participants with a CD19+ cell count greater than or equal to the lower limit of normal (LLN; reference range 0.11 to 0.66 giga [10^9] per liter) or the baseline value (whichever was lower) is presented. The baseline assessment is defined as the start of the Double-blind Period.
Time Frame: From baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 237 | 0
Participants
  TC 1, Week 8, n=0, 237, 0 |  | 1 |
  TC 1, Week 16, n=0, 182, 0 |  | 1 |
  TC 1, Week 24, n=0, 177, 0 |  | 2 |
  TC 1, Week 32, n=0, 96, 0 |  | 9 |
  TC 1, Week 40, n=0, 59, 0 |  | 3 |
  TC 1, Week 48, n=0, 46, 0 |  | 9 |
  TC 1, Week 56, n=0, 31, 0 |  | 5 |
  TC 1, Week 64, n=0, 23, 0 |  | 7 |
  TC 1, Week 72, n=0, 19, 0 |  | 4 |
  TC 1, Week 80, n=0, 15, 0 |  | 5 |
  TC 1, Week 88, n=0, 13, 0 |  | 1 |
  TC 1, Week 96, n=0, 12, 0 |  | 4 |
  TC 1, Week 104, n=0, 10, 0 |  | 1 |
  TC 1, Week 112, n=0, 8, 0 |  | 0 |
  TC 1, Week 120, n=0, 7, 0 |  | 1 |
  TC 1, Week 128, n=0, 4, 0 |  | 2 |
  TC 1, Week 136, n=0, 4, 0 |  | 1 |
  TC 1, Week 144, n=0, 4, 0 |  | 1 |
  TC 2, Week 8, n=0, 194, 0 |  | 1 |
  TC 2, Week 16, n=0, 177, 0 |  | 1 |
  TC 2, Week 24, n=0, 150, 0 |  | 1 |
  TC 2, Week 32, n=0, 97, 0 |  | 7 |
  TC 2, Week 40, n=0, 69, 0 |  | 12 |
  TC 2, Week 48, n=0, 58, 0 |  | 8 |
  TC 2, Week 56, n=0, 43, 0 |  | 13 |
  TC 2, Week 64, n=0, 31, 0 |  | 13 |
  TC 2, Week 72, n=0, 24, 0 |  | 11 |
  TC 2, Week 80, n=0, 21, 0 |  | 12 |
  TC 2, Week 88, n=0, 16, 0 |  | 7 |
  TC 2, Week 96, n=0, 10, 0 |  | 6 |
  TC 2, Week 104, n=0, 8, 0 |  | 5 |
  TC 2, Week 112, n=0, 4, 0 |  | 2 |
  TC 2, Week 120, n=0, 3, 0 |  | 2 |
  TC 2, Week 128, n=0, 1, 0 |  | 0 |
  TC 3, Week 8, n=0, 132, 0 |  | 0 |
  TC 3, Week 16, n=0, 119, 0 |  | 0 |
  TC 3, Week 24, n=0, 92, 0 |  | 0 |
  TC 3, Week 32, n=0, 63, 0 |  | 5 |
  TC 3, Week 40, n=0, 35, 0 |  | 4 |
  TC 3, Week 48, n=0, 24, 0 |  | 7 |
  TC 3, Week 56, n=0, 14, 0 |  | 2 |
  TC 3, Week 64, n=0, 10, 0 |  | 2 |
  TC 3, Week 72, n=0, 8, 0 |  | 5 |
  TC 3, Week 80, n=0, 8, 0 |  | 5 |
  TC 3, Week 88, n=0, 4, 0 |  | 3 |
  TC 3, Week 96, n=0, 2, 0 |  | 1 |
  TC 3, Week 104, n=0, 1, 0 |  | 1 |
  TC 4, Week 8, n=0, 70, 0 |  | 0 |
  TC 4, Week 16, n=0, 53, 0 |  | 0 |
  TC 4, Week 24, n=0, 37, 0 |  | 0 |
  TC 4, Week 32, n=0, 25, 0 |  | 4 |
  TC 4, Week 40, n=0, 8, 0 |  | 0 |
  TC 4, Week 48, n=0, 2, 0 |  | 1 |
  TC 5, Week 8, n=0, 30, 0 |  | 0 |
  TC 5, Week 16, n=0, 20, 0 |  | 0 |
  TC 5, Week 24, n=0, 20, 0 |  | 1 |
  TC 5, Week 32, n=0, 9, 0 |  | 2 |
  TC 5, Week 40, n=0, 3, 0 |  | 2 |
  TC 6, Week 8, n=0, 11, 0 |  | 0 |
  TC 6, Week 16, n=0, 10, 0 |  | 0 |
  TC 6, Week 24, n=0, 7, 0 |  | 0 |
  TC 6, Week 32, n=0, 2, 0 |  | 0 |
  TC 7, Week 8, n=0, 2, 0 |  | 0 |
  TC 7, Week 16, n=0, 1, 0 |  | 0 |

36. Secondary Outcome: Number of Participants With a CD3+ Cell Count Greater Than or Equal to the Lower Limit of Normal or the Baseline Value at the Indicated Time Point, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The number of participants with a CD3+ cell count greater than or equal to the lower limit of normal (LLN; reference range 0.11 to 0.66 giga [10^9] per liter) or the baseline value (whichever was lower) is presented. The baseline assessment is defined as the start of the Double-blind Period.
Time Frame: From baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 237 | 0
Participants
  TC 1, Week 8, n=0, 237, 0 |  | 197 |
  TC 1, Week 16, n=0, 182, 0 |  | 156 |
  TC 1, Week 24, n=0, 177, 0 |  | 152 |
  TC 1, Week 32, n=0, 96, 0 |  | 88 |
  TC 1, Week 40, n=0, 59, 0 |  | 51 |
  TC 1, Week 48, n=0, 46, 0 |  | 40 |
  TC 1, Week 56, n=0, 31, 0 |  | 26 |
  TC 1, Week 64, n=0, 23, 0 |  | 18 |
  TC 1, Week 72, n=0, 19, 0 |  | 16 |
  TC 1, Week 80, n=0, 15, 0 |  | 13 |
  TC 1, Week 88, n=0, 13, 0 |  | 11 |
  TC 1, Week 96, n=0, 12, 0 |  | 9 |
  TC 1, Week 104, n=0, 10, 0 |  | 9 |
  TC 1, Week 112, n=0, 8, 0 |  | 7 |
  TC 1, Week 120, n=0, 7, 0 |  | 6 |
  TC 1, Week 128, n=0, 4, 0 |  | 4 |
  TC 1, Week 136, n=0, 4, 0 |  | 4 |
  TC 1, Week 144, n=0, 4, 0 |  | 4 |
  TC 2, Week 8, n=0, 194, 0 |  | 170 |
  TC 2, Week 16, n=0, 177, 0 |  | 155 |
  TC 2, Week 24, n=0, 150, 0 |  | 128 |
  TC 2, Week 32, n=0, 97, 0 |  | 82 |
  TC 2, Week 40, n=0, 69, 0 |  | 60 |
  TC 2, Week 48, n=0, 58, 0 |  | 48 |
  TC 2, Week 56, n=0, 43, 0 |  | 35 |
  TC 2, Week 64, n=0, 31, 0 |  | 28 |
  TC 2, Week 72, n=0, 24, 0 |  | 20 |
  TC 2, Week 80, n=0, 21, 0 |  | 17 |
  TC 2, Week 88, n=0, 16, 0 |  | 14 |
  TC 2, Week 96, n=0, 10, 0 |  | 10 |
  TC 2, Week 104, n=0, 8, 0 |  | 8 |
  TC 2, Week 112, n=0, 4, 0 |  | 4 |
  TC 2, Week 120, n=0, 3, 0 |  | 3 |
  TC 2, Week 128, n=0, 1, 0 |  | 1 |
  TC 3, Week 8, n=0, 132, 0 |  | 118 |
  TC 3, Week 16, n=0, 119, 0 |  | 105 |
  TC 3, Week 24, n=0, 92, 0 |  | 81 |
  TC 3, Week 32, n=0, 63, 0 |  | 57 |
  TC 3, Week 40, n=0, 35, 0 |  | 32 |
  TC 3, Week 48, n=0, 24, 0 |  | 21 |
  TC 3, Week 56, n=0, 14, 0 |  | 12 |
  TC 3, Week 64, n=0, 10, 0 |  | 9 |
  TC 3, Week 72, n=0, 8, 0 |  | 8 |
  TC 3, Week 80, n=0, 8, 0 |  | 7 |
  TC 3, Week 88, n=0, 4, 0 |  | 4 |
  TC 3, Week 96, n=0, 2, 0 |  | 2 |
  TC 3, Week 104, n=0, 1, 0 |  | 1 |
  TC 4, Week 8, n=0, 70, 0 |  | 66 |
  TC 4, Week 16, n=0, 53, 0 |  | 49 |
  TC 4, Week 24, n=0, 37, 0 |  | 34 |
  TC 4, Week 32, n=0, 25, 0 |  | 23 |
  TC 4, Week 40, n=0, 8, 0 |  | 7 |
  TC 4, Week 48, n=0, 2, 0 |  | 2 |
  TC 5, Week 8, n=0, 30, 0 |  | 26 |
  TC 5, Week 16, n=0, 27, 0 |  | 24 |
  TC 5, Week 24, n=0, 20, 0 |  | 19 |
  TC 5, Week 32, n=0, 9, 0 |  | 9 |
  TC 5, Week 40, n=0, 3, 0 |  | 3 |
  TC 6, Week 8, n=0, 11, 0 |  | 9 |
  TC 6, Week 16, n=0, 10, 0 |  | 9 |
  TC 6, Week 24, n=0, 7, 0 |  | 6 |
  TC 6, Week 32, n=0, 2, 0 |  | 2 |
  TC 7, Week 8, n=0, 2, 0 |  | 2 |
  TC 7, Week 16, n=0, 1, 0 |  | 1 |

37. Secondary Outcome: Number of Participants With a CD4+ Cell Count Greater Than or Equal to the Lower Limit of Normal or the Baseline Value at the Indicated Time Point, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The number of participants with a CD4+ cell count greater than or equal to the lower limit of normal (LLN; reference range 0.11 to 0.66 giga [10^9] per liter) or the baseline value (whichever was lower) is presented. The baseline assessment is defined as the start of the Double-blind Period.
Time Frame: From baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 237 | 0
Participants
  TC 1, Week 8, n=0, 237, 0 |  | 209 |
  TC 1, Week 16, n=0, 182, 0 |  | 163 |
  TC 1, Week 24, n=0, 177, 0 |  | 150 |
  TC 1, Week 32, n=0, 96, 0 |  | 89 |
  TC 1, Week 40, n=0, 59, 0 |  | 50 |
  TC 1, Week 48, n=0, 46, 0 |  | 40 |
  TC 1, Week 56, n=0, 31, 0 |  | 26 |
  TC 1, Week 64, n=0, 23, 0 |  | 18 |
  TC 1, Week 72, n=0, 19, 0 |  | 16 |
  TC 1, Week 80, n=0, 15, 0 |  | 14 |
  TC 1, Week 88, n=0, 13, 0 |  | 10 |
  TC 1, Week 96, n=0, 12, 0 |  | 10 |
  TC 1, Week 104, n=0, 10, 0 |  | 9 |
  TC 1, Week 112, n=0, 8, 0 |  | 7 |
  TC 1, Week 120, n=0, 7, 0 |  | 6 |
  TC 1, Week 128, n=0, 4, 0 |  | 4 |
  TC 1, Week 136, n=0, 4, 0 |  | 4 |
  TC 1, Week 144, n=0, 4, 0 |  | 4 |
  TC 2, Week 8, n=0, 194, 0 |  | 174 |
  TC 2, Week 16, n=0, 177, 0 |  | 162 |
  TC 2, Week 24, n=0, 150, 0 |  | 136 |
  TC 2, Week 32, n=0, 97, 0 |  | 85 |
  TC 2, Week 40, n=0, 69, 0 |  | 63 |
  TC 2, Week 48, n=0, 58, 0 |  | 51 |
  TC 2, Week 56, n=0, 43, 0 |  | 37 |
  TC 2, Week 64, n=0, 31, 0 |  | 29 |
  TC 2, Week 72, n=0, 24, 0 |  | 22 |
  TC 2, Week 80, n=0, 21, 0 |  | 19 |
  TC 2, Week 88, n=0, 16, 0 |  | 15 |
  TC 2, Week 96, n=0, 10, 0 |  | 10 |
  TC 2, Week 104, n=0, 8, 0 |  | 8 |
  TC 2, Week 112, n=0, 4, 0 |  | 4 |
  TC 2, Week 120, n=0, 3, 0 |  | 3 |
  TC 2, Week 128, n=0, 1, 0 |  | 1 |
  TC 3, Week 8, n=0, 132, 0 |  | 120 |
  TC 3, Week 16, n=0, 119, 0 |  | 108 |
  TC 3, Week 24, n=0, 92, 0 |  | 81 |
  TC 3, Week 32, n=0, 63, 0 |  | 58 |
  TC 3, Week 40, n=0, 35, 0 |  | 33 |
  TC 3, Week 48, n=0, 24, 0 |  | 20 |
  TC 3, Week 56, n=0, 14, 0 |  | 13 |
  TC 3, Week 64, n=0, 10, 0 |  | 8 |
  TC 3, Week 72, n=0, 8, 0 |  | 8 |
  TC 3, Week 80, n=0, 8, 0 |  | 7 |
  TC 3, Week 88, n=0, 4, 0 |  | 4 |
  TC 3, Week 96, n=0, 2, 0 |  | 2 |
  TC 3, Week 104, n=0, 1, 0 |  | 1 |
  TC 4, Week 8, n=0, 70, 0 |  | 68 |
  TC 4, Week 16, n=0, 53, 0 |  | 51 |
  TC 4, Week 24, n=0, 37, 0 |  | 35 |
  TC 4, Week 32, n=0, 25, 0 |  | 24 |
  TC 4, Week 40, n=0, 8, 0 |  | 8 |
  TC 4, Week 48, n=0, 2, 0 |  | 2 |
  TC 5, Week 8, n=0, 30, 0 |  | 27 |
  TC 5, Week 16, n=0, 27, 0 |  | 26 |
  TC 5, Week 24, n=0, 20, 0 |  | 18 |
  TC 5, Week 32, n=0, 9, 0 |  | 9 |
  TC 5, Week 40, n=0, 3, 0 |  | 3 |
  TC 6, Week 8, n=0, 11, 0 |  | 10 |
  TC 6, Week 16, n=0, 10, 0 |  | 9 |
  TC 6, Week 24, n=0, 7, 0 |  | 7 |
  TC 6, Week 32, n=0, 2, 0 |  | 2 |
  TC 7, Week 8, n=0, 2, 0 |  | 2 |
  TC 7, Week 16, n=0, 1, 0 |  | 1 |

38. Secondary Outcome: Number of Participants With a CD8+ Cell Count Greater Than or Equal to the Lower Limit of Normal or the Baseline Value at the Indicated Time Point, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The number of participants with a CD8+ cell count greater than or equal to the lower limit of normal (LLN; reference range 0.11 to 0.66 giga [10^9] per liter) or the baseline value (whichever was lower) is presented. The baseline assessment is defined as the start of the Double-blind Period.
Time Frame: From baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 237 | 0
Participants
  TC 1, Week 8, n=0, 237, 0 |  | 216 |
  TC 1, Week 16, n=0, 182, 0 |  | 166 |
  TC 1, Week 24, n=0, 177, 0 |  | 160 |
  TC 1, Week 32, n=0, 96, 0 |  | 90 |
  TC 1, Week 40, n=0, 59, 0 |  | 51 |
  TC 1, Week 48, n=0, 46, 0 |  | 42 |
  TC 1, Week 56, n=0, 31, 0 |  | 29 |
  TC 1, Week 64, n=0, 23, 0 |  | 19 |
  TC 1, Week 72, n=0, 19, 0 |  | 15 |
  TC 1, Week 80, n=0, 15, 0 |  | 14 |
  TC 1, Week 88, n=0, 13, 0 |  | 12 |
  TC 1, Week 96, n=0, 12, 0 |  | 11 |
  TC 1, Week 104, n=0, 10, 0 |  | 10 |
  TC 1, Week 112, n=0, 8, 0 |  | 8 |
  TC 1, Week 120, n=0, 7, 0 |  | 6 |
  TC 1, Week 128, n=0, 4, 0 |  | 4 |
  TC 1, Week 136, n=0, 4, 0 |  | 4 |
  TC 1, Week 144, n=0, 4, 0 |  | 3 |
  TC 2, Week 8, n=0, 194, 0 |  | 181 |
  TC 2, Week 16, n=0, 177, 0 |  | 164 |
  TC 2, Week 24, n=0, 150, 0 |  | 140 |
  TC 2, Week 32, n=0, 97, 0 |  | 91 |
  TC 2, Week 40, n=0, 69, 0 |  | 65 |
  TC 2, Week 48, n=0, 58, 0 |  | 54 |
  TC 2, Week 56, n=0, 43, 0 |  | 40 |
  TC 2, Week 64, n=0, 31, 0 |  | 29 |
  TC 2, Week 72, n=0, 24, 0 |  | 23 |
  TC 2, Week 80, n=0, 21, 0 |  | 19 |
  TC 2, Week 88, n=0, 16, 0 |  | 15 |
  TC 2, Week 96, n=0, 10, 0 |  | 10 |
  TC 2, Week 104, n=0, 8, 0 |  | 8 |
  TC 2, Week 112, n=0, 4, 0 |  | 4 |
  TC 2, Week 120, n=0, 3, 0 |  | 3 |
  TC 2, Week 128, n=0, 1, 0 |  | 1 |
  TC 3, Week 8, n=0, 132, 0 |  | 128 |
  TC 3, Week 16, n=0, 119, 0 |  | 113 |
  TC 3, Week 24, n=0, 92, 0 |  | 88 |
  TC 3, Week 32, n=0, 63, 0 |  | 61 |
  TC 3, Week 40, n=0, 35, 0 |  | 34 |
  TC 3, Week 48, n=0, 24, 0 |  | 24 |
  TC 3, Week 56, n=0, 14, 0 |  | 13 |
  TC 3, Week 64, n=0, 10, 0 |  | 8 |
  TC 3, Week 72, n=0, 8, 0 |  | 8 |
  TC 3, Week 80, n=0, 8, 0 |  | 8 |
  TC 3, Week 88, n=0, 4, 0 |  | 4 |
  TC 3, Week 96, n=0, 2, 0 |  | 2 |
  TC 3, Week 104, n=0, 1, 0 |  | 1 |
  TC 4, Week 8, n=0, 70, 0 |  | 68 |
  TC 4, Week 16, n=0, 53, 0 |  | 52 |
  TC 4, Week 24, n=0, 37, 0 |  | 37 |
  TC 4, Week 32, n=0, 25, 0 |  | 24 |
  TC 4, Week 40, n=0, 8, 0 |  | 8 |
  TC 4, Week 48, n=0, 2, 0 |  | 2 |
  TC 5, Week 8, n=0, 30, 0 |  | 28 |
  TC 5, Week 16, n=0, 27, 0 |  | 26 |
  TC 5, Week 24, n=0, 20, 0 |  | 20 |
  TC 5, Week 32, n=0, 9, 0 |  | 9 |
  TC 5, Week 40, n=0, 3, 0 |  | 3 |
  TC 6, Week 8, n=0, 11, 0 |  | 10 |
  TC 6, Week 16, n=0, 10, 0 |  | 10 |
  TC 6, Week 24, n=0, 7, 0 |  | 6 |
  TC 6, Week 32, n=0, 2, 0 |  | 2 |
  TC 7, Week 8, n=0, 2, 0 |  | 2 |
  TC 7, Week 16, n=0, 1, 0 |  | 1 |

39. Secondary Outcome: Number of Participants With Vital Sign Data Outside the Clinical Concern Range at Baseline or Any Visit Post-baseline, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: The baseline value for a treatment course is defined as the value before infusion A of each treatment course. The post-baseline visit is defined as any assessment during or after the start of infusion A during the specified treatment course. Pre-defined limits of potential clinical concern for vital signs (Low, High) are: Diastolic blood pressure (DBP) (millimeters of mercury [mmHg]): 40, 110; Systolic blood pressure (SBP) (mmHg): 90, 170; Heart rate (beats per minute): 35, 120. LLN=lower limit of normal; ULN=upper limit of normal.
Time Frame: From baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 243 | 0
Participants
  DBP, TC 1, BL, <LLN, n=0, 242, 0 |  | 0 |
  DBP, TC 1, PBL, <LLN, n=0, 243, 0 |  | 2 |
  DBP, TC 1, BL, >ULN, n=0, 242, 0 |  | 1 |
  DBP, TC 1, PBL, >ULN, n=0, 243, 0 |  | 3 |
  SBP, TC 1, BL, <LLN, n=0, 242, 0 |  | 1 |
  SBP, TC 1, PBL, <LLN, n=0, 243, 0 |  | 15 |
  SBP, TC 1, BL, >ULN, n=0, 242, 0 |  | 1 |
  SBP, TC 1, PBL, >ULN, n=0, 243, 0 |  | 15 |
  HR, TC 1, BL, <LLN, n=0, 243, 0 |  | 0 |
  HR, TC 1, PBL, <LLN, n=0, 243, 0 |  | 0 |
  HR, TC 1, BL, >ULN, n=0, 243, 0 |  | 0 |
  HR, TC 1, PBL, >ULN, n=0, 243, 0 |  | 0 |
  DBP, TC 2, BL, <LLN, n=0, 196, 0 |  | 0 |
  DBP, TC 2, PBL, <LLN, n=0, 198, 0 |  | 0 |
  DBP, TC 2, BL, >ULN, n=0, 196, 0 |  | 0 |
  DBP, TC 2, PBL, >ULN, n=0, 198, 0 |  | 2 |
  SBP, TC 2, BL, <LLN, n=0, 196, 0 |  | 1 |
  SBP, TC 2, PBL, <LLN, n=0, 198, 0 |  | 9 |
  SBP, TC 2, BL, >ULN, n=0, 196, 0 |  | 0 |
  SBP, TC 2, PBL, >ULN, n=0, 198, 0 |  | 12 |
  HR, TC 2, BL, <LLN, n=0, 196, 0 |  | 0 |
  HR, TC 2, PBL, <LLN, n=0, 198, 0 |  | 0 |
  HR, TC 2, BL, >ULN, n=0, 196, 0 |  | 0 |
  HR, TC 2, PBL, >ULN, n=0, 198, 0 |  | 2 |
  DBP, TC 3, BL, <LLN, n=0, 136, 0 |  | 0 |
  DBP, TC 3, PBL, <LLN, n=0, 136, 0 |  | 1 |
  DBP, TC 3, BL, >ULN, n=0, 136, 0 |  | 0 |
  DBP, TC 3, PBL, >ULN, n=0, 136, 0 |  | 1 |
  SBP, TC 3, BL, <LLN, n=0, 136, 0 |  | 0 |
  SBP, TC 3, PBL, <LLN, n=0, 136, 0 |  | 6 |
  SBP, TC 3, BL, >ULN, n=0, 136, 0 |  | 1 |
  SBP, TC 3, PBL, >ULN, n=0, 136, 0 |  | 3 |
  HR, TC 3, BL, <LLN, n=0, 136, 0 |  | 0 |
  HR, TC 3, PBL, <LLN, n=0, 136, 0 |  | 0 |
  HR, TC 3, BL, >ULN, n=0, 136, 0 |  | 0 |
  HR, TC 3, PBL, >ULN, n=0, 136, 0 |  | 1 |
  DBP, TC 4, BL, <LLN, n=0, 72, 0 |  | 0 |
  DBP, TC 4, PBL, <LLN, n=0, 72, 0 |  | 0 |
  DBP, TC 4, BL, >ULN, n=0, 72, 0 |  | 0 |
  DBP, TC 4, PBL, >ULN, n=0, 72, 0 |  | 1 |
  SBP, TC 4, BL, <LLN, n=0, 72, 0 |  | 0 |
  SBP, TC 4, PBL, <LLN, n=0, 72, 0 |  | 4 |
  SBP, TC 4, BL, >ULN, n=0, 72, 0 |  | 0 |
  SBP, TC 4, PBL, >ULN, n=0, 72, 0 |  | 2 |
  HR, TC 4, BL, <LLN, n=0, 72, 0 |  | 0 |
  HR, TC 4, PBL, <LLN, n=0, 72, 0 |  | 0 |
  HR, TC 4, BL, >ULN, n=0, 72, 0 |  | 0 |
  HR, TC 4, PBL, >ULN, n=0, 72, 0 |  | 0 |
  DBP, TC 5, BL, <LLN, n=0, 31, 0 |  | 0 |
  DBP, TC 5, PBL, <LLN, n=0, 31, 0 |  | 0 |
  DBP, TC 5, BL, >ULN, n=0, 31, 0 |  | 0 |
  DBP, TC 5, PBL, >ULN, n=0, 31, 0 |  | 0 |
  SBP, TC 5, BL, <LLN, n=0, 31, 0 |  | 0 |
  SBP, TC 5, PBL, <LLN, n=0, 31, 0 |  | 1 |
  SBP, TC 5, BL, >ULN, n=0, 31, 0 |  | 0 |
  SBP, TC 5, PBL, >ULN, n=0, 31, 0 |  | 0 |
  HR, TC 5, BL, <LLN, n=0, 31, 0 |  | 0 |
  HR, TC 5, PBL, <LLN, n=0, 31, 0 |  | 0 |
  HR, TC 5, BL, >ULN, n=0, 31, 0 |  | 0 |
  HR, TC 5, PBL, >ULN, n=0, 31, 0 |  | 0 |
  DBP, TC 6, BL, <LLN, n=0, 11, 0 |  | 0 |
  DBP, TC 6, PBL, <LLN, n=0, 11, 0 |  | 0 |
  DBP, TC 6, BL, >ULN, n=0, 11, 0 |  | 0 |
  DBP, TC 6, PBL, >ULN, n=0, 11, 0 |  | 0 |
  SBP, TC 6, BL, <LLN, n=0, 11, 0 |  | 0 |
  SBP, TC 6, PBL, <LLN, n=0, 11, 0 |  | 0 |
  SBP, TC 6, BL, >ULN, n=0, 11, 0 |  | 0 |
  SBP, TC 6, PBL, >ULN, n=0, 11, 0 |  | 1 |
  HR, TC 6, BL, <LLN, n=0, 11, 0 |  | 0 |
  HR, TC 6, PBL, <LLN, n=0, 11, 0 |  | 0 |
  HR, TC 6, BL, >ULN, n=0, 11, 0 |  | 0 |
  HR, TC 6, PBL, >ULN, n=0, 11, 0 |  | 0 |
  DBP, TC 7, BL, <LLN, n=0, 2, 0 |  | 0 |
  DBP, TC 7, PBL, <LLN, n=0, 2, 0 |  | 0 |
  DBP, TC 7, BL, >ULN, n=0, 2, 0 |  | 0 |
  DBP, TC 7, PBL, >ULN, n=0, 2, 0 |  | 0 |
  SBP, TC 7, BL, <LLN, n=0, 2, 0 |  | 0 |
  SBP, TC 7, PBL, <LLN, n=0, 2, 0 |  | 0 |
  SBP, TC 7, BL, >ULN, n=0, 2, 0 |  | 0 |
  SBP, TC 7, PBL, >ULN, n=0, 2, 0 |  | 0 |
  HR, TC 7, BL, <LLN, n=0, 2, 0 |  | 0 |
  HR, TC 7, PBL, <LLN, n=0, 2, 0 |  | 0 |
  HR, TC 7, BL, >ULN, n=0, 2, 0 |  | 0 |
  HR, TC 7, PBL, >ULN, n=0, 2, 0 |  | 0 |

40. Secondary Outcome: Number of Participants With the Indicated Electrocardiogram (ECG) Findings, During the OL Period
Description: The number of participants with normal, abnormal clinically significant (CS), and abnormal not clinically significant (NCS) ECG findings, as well as the number of participants with no results (NR), during the OL Period are presented. An overall interpretation of the ECG was made by the investigator, or the investigator could delegate this task to a cardiologist, if applicable.
Time Frame: From DB Period completion (Week 24) until the completion of the OL Period, assessed up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 225 | 0
Participants
  Week 48, normal, n=0, 225, 0 |  | 150 |
  Week 48, abnormal CS, n=0, 225, 0 |  | 2 |
  Week 48, abnormal NCS, n=0, 225, 0 |  | 71 |
  Week 48, NR, n=0, 225, 0 |  | 2 |
  Week 72, normal, n=0, 202, 0 |  | 133 |
  Week 72, abnormal CS, n=0, 202, 0 |  | 1 |
  Week 72, abnormal NCS, n=0, 202, 0 |  | 67 |
  Week 72, NR, n=0, 202, 0 |  | 1 |
  Week 96, normal, n=0, 180, 0 |  | 119 |
  Week 96, abnormal CS, n=0, 180, 0 |  | 0 |
  Week 96, abnormal NCS, n=0, 180, 0 |  | 60 |
  Week 96, NR, n=0, 180, 0 |  | 1 |
  Week 120, normal, n=0, 167, 0 |  | 120 |
  Week 120, abnormal CS, n=0, 167, 0 |  | 1 |
  Week 120, abnormal NCS, n=0, 167, 0 |  | 46 |
  Week 120, NR, n=0, 167, 0 |  | 0 |
  Week 144, normal, n=0, 95, 0 |  | 68 |
  Week 144, abnormal CS, n=0, 95, 0 |  | 1 |
  Week 144, abnormal NCS, n=0, 95, 0 |  | 26 |
  Week 144, NR, n=0, 95, 0 |  | 0 |

41. Secondary Outcome: Number of Participants With the Indicated Clinical Chemistry Values of Potential Clinical Concern at Baseline or Any Visit Post-baseline, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: Only those parameters for which at least one value of clinical concern (CC) was reported are summarized. Baseline (BL) value for a treatment course (TC) is defined as the latest value on or before the date of infusion A of the TC. The post-baseline (PBL) visit is defined as any visit after the date of infusion A during the specified TC. Pre-defined limits of potential CC (CC Low [relative to the lower limit of normal], CC High [relative to the upper limit of normal]) are: Albumin: 0.9, 1.5; Alanine amino transferase (ALT): NA, 2; Alkaline phosphatase (ALP): NA, 1.5; Aspartate amino transferase (AST): NA, 2; Bilirubin total (TBIL): NA, 1.5; Calcium: 0.85, 1.08; CO2 content/bicarbonate (BCO): 0.85/0.75, 1.2/1.3, ; Chloride: 0.9, 1.1; Creatine kinase (CK): NA, 2; Creatinine: NA, 1.2; Gamma glutamyl transferase (GGT): NA, 2; Lactate dehydrogenase (LDH): NA, 2; Potassium: 0.9, 1.1; Sodium: 0.93, 1.07; Total protein: 0.8, 1.15; Urea/blood urea nitrogen (BUN): NA, 1.5; Uric acid: NA, 1.5.
Time Frame: From baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 239 | 0
Participants
  Albumin, TC 1, BL, CC low, n=0, 234, 0 |  | 0 |
  Albumin, TC 1, PBL, CC low, n=0, 239, 0 |  | 0 |
  ALT, TC 1, BL, CC high, n=0, 234, 0 |  | 0 |
  ALT, TC 1, PBL, CC high, n=0, 239, 0 |  | 3 |
  ALP, TC 1, BL, CC high, n=0, 234, 0 |  | 0 |
  ALP, TC 1, PBL, CC high, n=0, 239, 0 |  | 0 |
  AST, TC 1, BL, CC high, n=0, 234, 0 |  | 0 |
  AST, TC 1, PBL, CC high, n=0, 239, 0 |  | 1 |
  TBIL, TC 1, BL, CC high, n=0, 234, 0 |  | 0 |
  TBIL, TC 1, PBL, CC high, n=0, 239, 0 |  | 1 |
  Calcium, TC 1, BL, CC low, n=0, 234, 0 |  | 0 |
  Calcium, TC 1, PBL, CC low, n=0, 239, 0 |  | 1 |
  CO2/BCO, TC 1, BL, CC low, n=0, 234, 0 |  | 9 |
  CO2/BCO, TC 1, PBL, CC low, n=0, 239, 0 |  | 15 |
  Chloride, TC 1, BL, CC low, n=0, 234, 0 |  | 0 |
  Chloride, TC 1, PBL, CC low, n=0, 239, 0 |  | 0 |
  CK, TC 1, BL, CC high, n=0, 234, 0 |  | 1 |
  CK, TC 1, PBL, CC high, n=0, 239, 0 |  | 4 |
  Creatinine, TC 1, BL, CC high, n=0, 234, 0 |  | 0 |
  Creatinine, TC 1,PBL, CC high, n=0, 239, 0 |  | 0 |
  GGT, TC 1, BL, CC high, n=0, 234, 0 |  | 11 |
  GGT, TC 1, PBL, CC high, n=0, 239, 0 |  | 9 |
  LDH, TC 1, BL, CC high, n=0, 234, 0 |  | 1 |
  LDH, TC 1, PBL, CC high, n=0, 239, 0 |  | 1 |
  Potassium, TC 1, BL, CC high, n=0, 234, 0 |  | 2 |
  Potassium, TC 1, PBL, CC high, n=0, 239, 0 |  | 2 |
  Potassium, TC 1, BL, CC low, n=0, 234, 0 |  | 0 |
  Potassium, TC 1, PBL, CC low, n=0, 239, 0 |  | 0 |
  Sodium, TC 1, BL, CC low, n=0, 234, 0 |  | 0 |
  Sodium, TC 1, PBL, CC low, n=0, 239, 0 |  | 1 |
  Total Protein, TC 1, BL, CC low, n=0, 234, 0 |  | 0 |
  Total Protein, TC 1, PBL, CC low, n=0, 239, 0 |  | 0 |
  Urea/BUN, TC 1, BL, CC high, n=0, 234, 0 |  | 0 |
  Urea/BUN, TC 1, PBL, CC high, n=0, 239, 0 |  | 1 |
  Uric acid, TC 1, BL, CC high, n=0, 234, 0 |  | 0 |
  Uric acid, TC 1, PBL, CC high, n=0, 239, 0 |  | 0 |
  Albumin, TC 2, BL, CC low, n=0, 177, 0 |  | 1 |
  Albumin, TC 2, PBL, CC low, n=0, 196, 0 |  | 0 |
  ALT, TC 2, BL, CC high, n=0, 177, 0 |  | 0 |
  ALT, TC 2, PBL, CC high, n=0, 196, 0 |  | 2 |
  ALP, TC 2, BL, CC high, n=0, 177, 0 |  | 1 |
  ALP, TC 2, PBL, CC high, n=0, 196, 0 |  | 1 |
  AST, TC 2, BL, CC high, n=0, 176, 0 |  | 0 |
  AST, TC 2, PBL, CC high, n=0, 196, 0 |  | 1 |
  TBIL, TC 2, BL, CC high, n=0, 177, 0 |  | 0 |
  TBIL, TC 2, PBL, CC high, n=0, 196, 0 |  | 1 |
  Calcium, TC 2, BL, CC low, n=0, 176, 0 |  | 1 |
  Calcium, TC 2, PBL, CC low, n=0, 196, 0 |  | 0 |
  CO2/BCO, TC 2, BL, CC low, n=0, 176, 0 |  | 5 |
  CO2/BCO, TC 2, PBL, CC low, n=0, 196, 0 |  | 10 |
  Chloride, TC 2, BL, CC low, n=0, 177, 0 |  | 0 |
  Chloride, TC 2, PBL, CC low, n=0, 196, 0 |  | 1 |
  CK, TC 2, BL, CC high, n=0, 177, 0 |  | 0 |
  CK, TC 2, PBL, CC high, n=0, 196, 0 |  | 4 |
  Creatinine, TC 2, BL, CC high, n=0, 177, 0 |  | 1 |
  Creatinine, TC 2,PBL, CC high, n=0, 196, 0 |  | 0 |
  GGT, TC 2, BL, CC high, n=0, 117, 0 |  | 3 |
  GGT, TC 2, PBL, CC high, n=0, 196, 0 |  | 9 |
  LDH, TC 2, BL, CC high, n=0, 176, 0 |  | 0 |
  LDH, TC 2, PBL, CC high, n=0, 196, 0 |  | 0 |
  Potassium, TC 2, BL, CC high, n=0, 176, 0 |  | 1 |
  Potassium, TC 2, PBL, CC high, n=0, 196, 0 |  | 1 |
  Potassium, TC 2, BL, CC low, n=0, 176, 0 |  | 1 |
  Potassium, TC 2, PBL, CC low, n=0, 196, 0 |  | 1 |
  Sodium, TC 2, BL, CC low, n=0, 177, 0 |  | 0 |
  Sodium, TC 2, PBL, CC low, n=0, 196, 0 |  | 1 |
  Total Protein, TC 2, BL, CC low, n=0, 177, 0 |  | 1 |
  Total Protein, TC 2, PBL, CC low, n=0, 196, 0 |  | 0 |
  Urea/BUN, TC 2, BL, CC high, n=0, 177, 0 |  | 1 |
  Urea/BUN, TC 2, PBL, CC high, n=0, 196, 0 |  | 1 |
  Uric acid, TC 2, BL, CC high, n=0, 177, 0 |  | 0 |
  Uric acid, TC 2, PBL, CC high, n=0, 196, 0 |  | 0 |
  Albumin, TC 3, BL, CC low, n=0, 116, 0 |  | 0 |
  Albumin, TC 3, PBL, CC low, n=0, 134, 0 |  | 0 |
  ALT, TC 3, BL, CC high, n=0, 116, 0 |  | 1 |
  ALT, TC 3, PBL, CC high, n=0, 135, 0 |  | 2 |
  ALP, TC 3, BL, CC high, n=0, 116, 0 |  | 1 |
  ALP, TC 3, PBL, CC high, n=0, 135, 0 |  | 3 |
  AST, TC 3, BL, CC high, n=0, 116, 0 |  | 0 |
  AST, TC 3, PBL, CC high, n=0, 135, 0 |  | 2 |
  TBIL, TC 3, BL, CC high, n=0, 116, 0 |  | 0 |
  TBIL, TC 3, PBL, CC high, n=0, 135, 0 |  | 1 |
  Calcium, TC 3, BL, CC low, n=0, 116, 0 |  | 0 |
  Calcium, TC 3, PBL, CC low, n=0, 134, 0 |  | 1 |
  CO2/BCO, TC 3, BL, CC low, n=0, 116, 0 |  | 2 |
  CO2/BCO, TC 3, PBL, CC low, n=0, 134, 0 |  | 6 |
  Chloride, TC 3, BL, CC low, n=0, 116, 0 |  | 0 |
  Chloride, TC 3, PBL, CC low, n=0, 134, 0 |  | 0 |
  CK, TC 3, BL, CC high, n=0, 116, 0 |  | 2 |
  CK, TC 3, PBL, CC high, n=0, 135, 0 |  | 2 |
  Creatinine, TC 3, BL, CC high, n=0, 116, 0 |  | 0 |
  Creatinine, TC 3, PBL, CC high, n=0, 134, 0 |  | 1 |
  GGT, TC 3, BL, CC high, n=0, 116, 0 |  | 5 |
  GGT, TC 3, PBL, CC high, n=0, 134, 0 |  | 7 |
  LDH, TC 3, BL, CC high, n=0, 116, 0 |  | 0 |
  LDH, TC 3, PBL, CC high, n=0, 135, 0 |  | 1 |
  Potassium, TC 3, BL, CC high, n=0, 116, 0 |  | 0 |
  Potassium, TC 3, PBL, CC high, n=0, 134, 0 |  | 0 |
  Potassium, TC 3, BL, CC low, n=0, 116, 0 |  | 0 |
  Potassium, TC 3, PBL, CC low, n=0, 134, 0 |  | 2 |
  Sodium, TC 3, BL, CC low, n=0, 116, 0 |  | 0 |
  Sodium, TC 3, PBL, CC low, n=0, 134, 0 |  | 0 |
  Total Protein, TC 3, BL, CC low, n=0, 116, 0 |  | 0 |
  Total Protein, TC 3, PBL, CC low, n=0, 134, 0 |  | 0 |
  Urea/BUN, TC 3, BL, CC high, n=0, 116, 0 |  | 1 |
  Urea/BUN, TC 3, PBL, CC high, n=0, 134, 0 |  | 1 |
  Uric acid, TC 3, BL, CC high, n=0, 116, 0 |  | 0 |
  Uric acid, TC 3, PBL, CC high, n=0, 134, 0 |  | 1 |
  Albumin, TC 4, BL, CC low, n=0, 67, 0 |  | 0 |
  Albumin, TC 4, PBL, CC low, n=0, 72, 0 |  | 0 |
  ALT, TC 4, BL, CC high, n=0, 67, 0 |  | 1 |
  ALT, TC 4, PBL, CC high, n=0, 72, 0 |  | 2 |
  ALP, TC 4, BL, CC high, n=0, 67, 0 |  | 0 |
  ALP, TC 4, PBL, CC high, n=0, 72, 0 |  | 1 |
  AST, TC 4, BL, CC high, n=0, 67, 0 |  | 1 |
  AST, TC 4, PBL, CC high, n=0, 72, 0 |  | 2 |
  TBIL, TC 4, BL, CC high, n=0, 67, 0 |  | 0 |
  TBIL, TC 4, PBL, CC high, n=0, 72, 0 |  | 0 |
  Calcium, TC 4, BL, CC low, n=0, 67, 0 |  | 0 |
  Calcium, TC 4, PBL, CC low, n=0, 72, 0 |  | 0 |
  CO2/BCO, TC 4, BL, CC low, n=0, 67, 0 |  | 1 |
  CO2/BCO, TC 4, PBL, CC low, n=0, 72, 0 |  | 2 |
  Chloride, TC 4, BL, CC low, n=0, 67, 0 |  | 0 |
  Chloride, TC 4, PBL, CC low, n=0, 72, 0 |  | 0 |
  CK, TC 4, BL, CC high, n=0, 67, 0 |  | 0 |
  CK, TC 4, PBL, CC high, n=0, 72, 0 |  | 1 |
  Creatinine, TC 4, BL, CC high, n=0, 67, 0 |  | 1 |
  Creatinine, TC 4, PBL, CC high, n=0, 72, 0 |  | 1 |
  GGT, TC 4, BL, CC high, n=0, 67, 0 |  | 2 |
  GGT, TC 4, PBL, CC high, n=0, 72, 0 |  | 3 |
  LDH, TC 4, BL, CC high, n=0, 67, 0 |  | 0 |
  LDH, TC 4, PBL, CC high, n=0, 72, 0 |  | 0 |
  Potassium, TC 4, BL, CC high, n=0, 67, 0 |  | 0 |
  Potassium, TC 4, PBL, CC high, n=0, 72, 0 |  | 0 |
  Potassium, TC 4, BL, CC low, n=0, 67, 0 |  | 0 |
  Potassium, TC 4, PBL, CC low, n=0, 72, 0 |  | 0 |
  Sodium, TC 4, BL, CC low, n=0, 67, 0 |  | 0 |
  Sodium, TC 4, PBL, CC low, n=0, 72, 0 |  | 0 |
  Total Protein, TC 4, BL, CC low, n=0, 67, 0 |  | 0 |
  Total Protein, TC 4, PBL, CC low, n=0, 72, 0 |  | 0 |
  Urea/BUN, TC 4, BL, CC high, n=0, 67, 0 |  | 0 |
  Urea/BUN, TC 4, PBL, CC high, n=0, 72, 0 |  | 1 |
  Uric acid, TC 4, BL, CC high, n=0, 67, 0 |  | 0 |
  Uric acid, TC 4, PBL, CC high, n=0, 72, 0 |  | 0 |
  Albumin, TC 5, BL, CC low, n=0, 29, 0 |  | 0 |
  Albumin, TC 5, PBL, CC low, n=0, 31, 0 |  | 0 |
  ALT, TC 5, BL, CC high, n=0, 29, 0 |  | 0 |
  ALT, TC 5, PBL, CC high, n=0, 31, 0 |  | 1 |
  ALP, TC 5, BL, CC high, n=0, 29, 0 |  | 0 |
  ALP, TC 5, PBL, CC high, n=0, 31, 0 |  | 1 |
  AST, TC 5, BL, CC high, n=0, 29, 0 |  | 0 |
  AST, TC 5, PBL, CC high, n=0, 31, 0 |  | 0 |
  TBIL, TC 5, BL, CC high, n=0, 29, 0 |  | 0 |
  TBIL, TC 3, PBL, CC high, n=0, 31, 0 |  | 0 |
  Calcium, TC 5, BL, CC low, n=0, 29, 0 |  | 0 |
  Calcium, TC 5, PBL, CC low, n=0, 31, 0 |  | 0 |
  CO2/BCO, TC 5, BL, CC low, n=0, 29, 0 |  | 0 |
  CO2/BCO, TC 5, PBL, CC low, n=0, 31, 0 |  | 0 |
  Chloride, TC 5, BL, CC low, n=0, 29, 0 |  | 0 |
  Chloride, TC 5, PBL, CC low, n=0, 31, 0 |  | 0 |
  CK, TC 5, BL, CC high, n=0, 29, 0 |  | 0 |
  CK, TC 5, PBL, CC high, n=0, 31, 0 |  | 1 |
  Creatinine, TC 5, BL, CC high, n=0, 29, 0 |  | 0 |
  Creatinine, TC 5, PBL, CC high, n=0, 31, 0 |  | 0 |
  GGT, TC 5, BL, CC high, n=0, 29, 0 |  | 0 |
  GGT, TC 5, PBL, CC high, n=0, 31, 0 |  | 1 |
  LDH, TC 5, BL, CC high, n=0, 29, 0 |  | 0 |
  LDH, TC 5, PBL, CC high, n=0, 31, 0 |  | 0 |
  Potassium, TC 5, BL, CC high, n=0, 29, 0 |  | 0 |
  Potassium, TC 5, PBL, CC high, n=0, 31, 0 |  | 0 |
  Potassium, TC 5, BL, CC low, n=0, 29, 0 |  | 0 |
  Potassium, TC 5, PBL, CC low, n=0, 31, 0 |  | 0 |
  Sodium, TC 5, BL, CC low, n=0, 29, 0 |  | 0 |
  Sodium, TC 5, PBL, CC low, n=0, 31, 0 |  | 0 |
  Total Protein, TC 5, BL, CC low, n=0, 29, 0 |  | 0 |
  Total Protein, TC 5, PBL, CC low, n=0, 31, 0 |  | 0 |
  Urea/BUN, TC 5, BL, CC high, n=0, 29, 0 |  | 0 |
  Urea/BUN, TC 5, PBL, CC high, n=0, 31, 0 |  | 0 |
  Uric acid, TC 5, BL, CC high, n=0, 29, 0 |  | 0 |
  Uric acid, TC 5, PBL, CC high, n=0, 31, 0 |  | 0 |
  Albumin, TC 6, BL, CC low, n=0, 11, 0 |  | 0 |
  Albumin, TC 6, PBL, CC low, n=0, 11, 0 |  | 0 |
  ALT, TC 6, BL, CC high, n=0, 11, 0 |  | 0 |
  ALT, TC 6, PBL, CC high, n=0, 11, 0 |  | 0 |
  ALP, TC 6, BL, CC high, n=0, 11, 0 |  | 0 |
  ALP, TC 6, PBL, CC high, n=0, 11, 0 |  | 0 |
  AST, TC 6, BL, CC high, n=0, 10, 0 |  | 0 |
  AST, TC 6, PBL, CC high, n=0, 11, 0 |  | 0 |
  TBIL, TC 6, BL, CC high, n=0, 11, 0 |  | 0 |
  TBIL, TC 6, PBL, CC high, n=0, 11, 0 |  | 0 |
  Calcium, TC 6, BL, CC low, n=0, 10, 0 |  | 0 |
  Calcium, TC 6, PBL, CC low, n=0, 11, 0 |  | 0 |
  CO2/BCO, TC 6, BL, CC low, n=0, 10, 0 |  | 0 |
  CO2/BCO, TC 6, PBL, CC low, n=0, 11, 0 |  | 1 |
  Chloride, TC 6, BL, CC low, n=0, 11, 0 |  | 0 |
  Chloride, TC 6, PBL, CC low, n=0, 11, 0 |  | 0 |
  CK, TC 6, BL, CC high, n=0, 11, 0 |  | 0 |
  CK, TC 6, PBL, CC high, n=0, 11, 0 |  | 0 |
  Creatinine, TC 6, BL, CC high, n=0, 11, 0 |  | 0 |
  Creatinine, TC 6, PBL, CC high, n=0, 11, 0 |  | 0 |
  GGT, TC 6, BL, CC high, n=0, 11, 0 |  | 0 |
  GGT, TC 6, PBL, CC high, n=0, 11, 0 |  | 0 |
  LDH, TC 6, BL, CC high, n=0, 10, 0 |  | 0 |
  LDH, TC 6, PBL, CC high, n=0, 11, 0 |  | 0 |
  Potassium, TC 6, BL, CC high, n=0, 10, 0 |  | 0 |
  Potassium, TC 6, PBL, CC high, n=0, 11, 0 |  | 0 |
  Potassium, TC 6, BL, CC low, n=0, 10, 0 |  | 0 |
  Potassium, TC 6, PBL, CC low, n=0, 11, 0 |  | 0 |
  Sodium, TC 6, BL, CC low, n=0, 11, 0 |  | 0 |
  Sodium, TC 6, PBL, CC low, n=0, 11, 0 |  | 0 |
  Total Protein, TC 6, BL, CC low, n=0, 11, 0 |  | 0 |
  Total Protein, TC 6, PBL, CC low, n=0, 11, 0 |  | 0 |
  Urea/BUN, TC 6, BL, CC high, n=0, 11, 0 |  | 0 |
  Urea/BUN, TC 6, PBL, CC high, n=0, 11, 0 |  | 0 |
  Uric acid, TC 6, BL, CC high, n=0, 11, 0 |  | 0 |
  Uric acid, TC 6, PBL, CC high, n=0, 11, 0 |  | 0 |
  Albumin, TC 7, BL, CC low, n=0, 2, 0 |  | 0 |
  Albumin, TC 7, PBL, CC low, n=0, 2, 0 |  | 0 |
  ALT, TC 7, BL, CC high, n=0, 2, 0 |  | 0 |
  ALT, TC 7, PBL, CC high, n=0, 2, 0 |  | 0 |
  ALP, TC 7, BL, CC high, n=0, 2, 0 |  | 0 |
  ALP, TC 7, PBL, CC high, n=0, 2, 0 |  | 0 |
  AST, TC 7, BL, CC high, n=0, 2, 0 |  | 0 |
  AST, TC 7, PBL, CC high, n=0, 2, 0 |  | 0 |
  TBIL, TC 7, BL, CC high, n=0, 2, 0 |  | 0 |
  TBIL, TC 7, PBL, CC high, n=0, 2, 0 |  | 0 |
  Calcium, TC 7, BL, CC low, n=0, 2, 0 |  | 0 |
  Calcium, TC 7, PBL, CC low, n=0, 2, 0 |  | 0 |
  CO2/BCO, TC 7, BL, CC low, n=0, 2, 0 |  | 0 |
  CO2/BCO, TC 7, PBL, CC low, n=0, 2, 0 |  | 0 |
  Chloride, TC 7, BL, CC low, n=0, 2, 0 |  | 0 |
  Chloride, TC 7, PBL, CC low, n=0, 2, 0 |  | 0 |
  CK, TC 7, BL, CC high, n=0, 2, 0 |  | 0 |
  CK, TC 7, PBL, CC high, n=0, 2, 0 |  | 0 |
  Creatinine, TC 7, BL, CC high, n=0, 2, 0 |  | 0 |
  Creatinine, TC 7, PBL, CC high, n=0, 2, 0 |  | 0 |
  GGT, TC 7, BL, CC high, n=0, 2, 0 |  | 0 |
  GGT, TC 7, PBL, CC high, n=0, 2, 0 |  | 0 |
  LDH, TC 7, BL, CC high, n=0, 2, 0 |  | 0 |
  LDH, TC 7, PBL, CC high, n=0, 2, 0 |  | 0 |
  Potassium, TC 7, BL, CC high, n=0, 2, 0 |  | 0 |
  Potassium, TC 7, PBL, CC high, n=0, 2, 0 |  | 0 |
  Potassium, TC 7, BL, CC low, n=0, 2, 0 |  | 0 |
  Potassium, TC 7, PBL, CC low, n=0, 2, 0 |  | 0 |
  Sodium, TC 7, BL, CC low, n=0, 2, 0 |  | 0 |
  Sodium, TC 7, PBL, CC low, n=0, 2, 0 |  | 0 |
  Total Protein, TC 7, BL, CC low, n=0, 2, 0 |  | 0 |
  Total Protein, TC 7, PBL, CC low, n=0, 2, 0 |  | 0 |
  Urea/BUN, TC 7, BL, CC high, n=0, 2, 0 |  | 0 |
  Urea/BUN, TC 7, PBL, CC high, n=0, 2, 0 |  | 0 |
  Uric acid, TC 7, BL, CC high, n=0, 2, 0 |  | 0 |
  Uric acid, TC 7, PBL, CC high, n=0, 2, 0 |  | 0 |

42. Secondary Outcome: Number of Participants With the Indicated Hematology Values of Potential Clinical Concern at Baseline or Any Visit Post-baseline, During the DB and OL Periods, by Ofatumumab Treatment Course
Description: Only those parameters for which at least one value of clinical concern (CC) was reported are summarized. The baseline (BL) value for a treatment course (TC) is defined as the latest value on or before the date of infusion A of the TC. The post-baseline (PBL) visit is defined as any visit after the date of infusion A during the specified TC. Pre-defined limits of potential clinical concern (CC Low [relative to lower limit of normal], CC High [relative to upper limit of normal]) are: Eosinophils: NA, 2; Hematocrit (HCT): 0.75, 1.2; Hemoglobin (Hb): 0.75, 1.2; Lymphocytes: 0.4, 2; Neutrophils total (TNUE): 0.8, 1.6; Platelet count (PC): 0.65, 1.5; Red blood cell count (RBC): 0.75, 2; White blood cell count (WBC): 0.7, 1.6.
Time Frame: From baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 239 | 0
Participants
  Eosinophils, TC 1, BL, CC high, n=0, 224, 0 |  | 2 |
  Eosinophils, TC 1, PBL, CC high, n=0, 239, 0 |  | 4 |
  HCT, TC 1, BL, CC low, n=0, 224, 0 |  | 0 |
  HCT, TC 1, PBL, CC low, n=0, 239, 0 |  | 2 |
  Hb, TC 1, BL, CC low, n=0, 224, 0 |  | 3 |
  Hb, TC 1, PBL, CC low, n=0, 239, 0 |  | 6 |
  Lymphocytes, TC 1, BL, CC low, n=0, 232, 0 |  | 1 |
  Lymphocytes, TC 1, PBL, CC low, n=0, 239, 0 |  | 1 |
  PC, TC 1, BL, CC high, n=0, 221, 0 |  | 1 |
  PC, TC 1, PBL, CC high, n=0, 239, 0 |  | 3 |
  RBC count, TC 1, BL, CC low, n=0, 224, 0 |  | 1 |
  RBC count, TC 1, PBL, CC low, n=0, 239, 0 |  | 1 |
  TNUE, TC 1, BL, CC low, n=0, 224, 0 |  | 0 |
  TNUE, TC 1, PBL, CC low, n=0, 239, 0 |  | 8 |
  TNUE, TC 1, BL, CC high, n=0, 224, 0 |  | 5 |
  TNUE, TC 1,PBL, CC high, n=0, 239, 0 |  | 6 |
  WBC count, TC 1, BL, CC low, n=0, 224, 0 |  | 0 |
  WBC count, TC 1, PBL, CC low, n=0, 239, 0 |  | 1 |
  WBC count, TC 1, BL, CC high, n=0, 224, 0 |  | 1 |
  WBC count, TC 1, PBL, CC high, n=0, 239, 0 |  | 1 |
  Eosinophils, TC 2, BL, CC high, n=0, 171, 0 |  | 2 |
  Eosinophils, TC 2, PBL, CC high, n=0, 195, 0 |  | 6 |
  HCT, TC 2, BL, CC low, n=0, 173, 0 |  | 0 |
  HCT, TC 2, PBL, CC low, n=0, 195, 0 |  | 0 |
  Hb, TC 2, BL, CC low, n=0, 172, 0 |  | 0 |
  Hb, TC 2, PBL, CC low, n=0, 195, 0 |  | 1 |
  Lymphocytes, TC 2, BL, CC low, n=0, 177, 0 |  | 0 |
  Lymphocytes, TC 2, PBL, CC low, n=0, 196, 0 |  | 1 |
  PC, TC 2, BL, CC high, n=0, 170, 0 |  | 0 |
  PC, TC 2, PBL, CC high, n=0, 195, 0 |  | 0 |
  RBC count, TC 2, BL, CC low, n=0, 172, 0 |  | 0 |
  RBC count, TC 2, PBL, CC low, n=0, 195, 0 |  | 0 |
  TNUE, TC 2, BL, CC low, n=0, 171, 0 |  | 1 |
  TNUE, TC 2, PBL, CC low, n=0, 195, 0 |  | 3 |
  TNUE, TC 2, BL, CC high, n=0, 171, 0 |  | 0 |
  TNUE, TC 2,PBL, CC high, n=0, 195, 0 |  | 1 |
  WBC count, TC 2, BL, CC low, n=0, 171, 0 |  | 1 |
  WBC count, TC 2, PBL, CC low, n=0, 195, 0 |  | 1 |
  WBC count, TC 2, BL, CC high, n=0, 171, 0 |  | 0 |
  WBC count, TC 2, PBL, CC high, n=0, 195, 0 |  | 1 |
  Eosinophils, TC 3, BL, CC high, n=0, 114, 0 |  | 2 |
  Eosinophils, TC 3, PBL, CC high, n=0, 134, 0 |  | 2 |
  HCT, TC 3, BL, CC low, n=0, 115, 0 |  | 0 |
  HCT, TC 3, PBL, CC low, n=0, 134, 0 |  | 0 |
  Hb, TC 3, BL, CC low, n=0, 115, 0 |  | 0 |
  Hb, TC 3, PBL, CC low, n=0, 134, 0 |  | 0 |
  Lymphocytes, TC 3, BL, CC low, n=0, 117, 0 |  | 0 |
  Lymphocytes, TC 3, PBL, CC low, n=0, 134, 0 |  | 0 |
  PC, TC 3, BL, CC high, n=0, 115, 0 |  | 0 |
  PC, TC 3, PBL, CC high, n=0, 134, 0 |  | 0 |
  RBC count, TC 3, BL, CC low, n=0, 115, 0 |  | 0 |
  RBC count, TC 3, PBL, CC low, n=0, 134, 0 |  | 0 |
  TNUE, TC 3, BL, CC low, n=0, 114, 0 |  | 0 |
  TNUE, TC 3, PBL, CC low, n=0, 134, 0 |  | 2 |
  TNUE, TC 3, BL, CC high, n=0, 114, 0 |  | 0 |
  TNUE, TC 3,PBL, CC high, n=0, 134, 0 |  | 0 |
  WBC count, TC 3, BL, CC low, n=0, 114, 0 |  | 0 |
  WBC count, TC 3, PBL, CC low, n=0, 134, 0 |  | 0 |
  WBC count, TC 3, BL, CC high, n=0, 114, 0 |  | 0 |
  WBC count, TC 3, PBL, CC high, n=0, 134, 0 |  | 0 |
  Eosinophils, TC 4, BL, CC high, n=0, 66, 0 |  | 1 |
  Eosinophils, TC 4, PBL, CC high, n=0, 72, 0 |  | 1 |
  HCT, TC 4, BL, CC low, n=0, 66, 0 |  | 0 |
  HCT, TC 4, PBL, CC low, n=0, 72, 0 |  | 0 |
  Hb, TC 4, BL, CC low, n=0, 66, 0 |  | 0 |
  Hb, TC 4, PBL, CC low, n=0, 72, 0 |  | 0 |
  Lymphocytes, TC 4, BL, CC low, n=0, 67, 0 |  | 0 |
  Lymphocytes, TC 4, PBL, CC low, n=0, 72, 0 |  | 0 |
  PC, TC 4, BL, CC high, n=0, 65, 0 |  | 0 |
  PC, TC 4, PBL, CC high, n=0, 72, 0 |  | 0 |
  RBC count, TC 4, BL, CC low, n=0, 66, 0 |  | 0 |
  RBC count, TC 4, PBL, CC low, n=0, 72, 0 |  | 0 |
  TNUE, TC 4, BL, CC low, n=0, 66, 0 |  | 0 |
  TNUE, TC 4, PBL, CC low, n=0, 72, 0 |  | 5 |
  TNUE, TC 4, BL, CC high, n=0, 66, 0 |  | 0 |
  TNUE, TC 4,PBL, CC high, n=0, 72, 0 |  | 0 |
  WBC count, TC 4, BL, CC low, n=0, 66, 0 |  | 0 |
  WBC count, TC 4, PBL, CC low, n=0, 72, 0 |  | 0 |
  WBC count, TC 4, BL, CC high, n=0, 66, 0 |  | 0 |
  WBC count, TC 4, PBL, CC high, n=0, 72, 0 |  | 0 |
  Eosinophils, TC 5, BL, CC high, n=0, 29, 0 |  | 0 |
  Eosinophils, TC 5, PBL, CC high, n=0, 31, 0 |  | 1 |
  HCT, TC 5, BL, CC low, n=0, 29, 0 |  | 0 |
  HCT, TC 5, PBL, CC low, n=0, 31, 0 |  | 0 |
  Hb, TC 5, BL, CC low, n=0, 29, 0 |  | 0 |
  Hb, TC 5, PBL, CC low, n=0, 31, 0 |  | 0 |
  Lymphocytes, TC 5, BL, CC low, n=0, 29, 0 |  | 0 |
  Lymphocytes, TC 5, PBL, CC low, n=0, 31, 0 |  | 0 |
  PC, TC 5, BL, CC high, n=0, 29, 0 |  | 0 |
  PC, TC 5, PBL, CC high, n=0, 31, 0 |  | 0 |
  RBC count, TC 5, BL, CC low, n=0, 29, 0 |  | 0 |
  RBC count, TC 5, PBL, CC low, n=0, 31, 0 |  | 0 |
  TNUE, TC 5, BL, CC low, n=0, 29, 0 |  | 2 |
  TNUE, TC 5, PBL, CC low, n=0, 31, 0 |  | 0 |
  TNUE, TC 5, BL, CC high, n=0, 29, 0 |  | 0 |
  TNUE, TC 5,PBL, CC high, n=0, 31, 0 |  | 0 |
  WBC count, TC 5, BL, CC low, n=0, 29, 0 |  | 0 |
  WBC count, TC 5, PBL, CC low, n=0, 31, 0 |  | 0 |
  WBC count, TC 5, BL, CC high, n=0, 29, 0 |  | 0 |
  WBC count, TC 5, PBL, CC high, n=0, 31, 0 |  | 0 |
  Eosinophils, TC 6, BL, CC high, n=0, 11, 0 |  | 0 |
  Eosinophils, TC 6, PBL, CC high, n=0, 11, 0 |  | 0 |
  HCT, TC 6, BL, CC low, n=0, 11, 0 |  | 0 |
  HCT, TC 6, PBL, CC low, n=0, 11, 0 |  | 0 |
  Hb, TC 6, BL, CC low, n=0, 11, 0 |  | 1 |
  Hb, TC 6, PBL, CC low, n=0, 11, 0 |  | 0 |
  Lymphocytes, TC 6, BL, CC low, n=0, 11, 0 |  | 0 |
  Lymphocytes, TC 6, PBL, CC low, n=0, 11, 0 |  | 0 |
  PC, TC 6, BL, CC high, n=0, 11, 0 |  | 0 |
  PC, TC 6, PBL, CC high, n=0, 11, 0 |  | 0 |
  RBC count, TC 6, BL, CC low, n=0, 11, 0 |  | 0 |
  RBC count, TC 6, PBL, CC low, n=0, 11, 0 |  | 0 |
  TNUE, TC 6, BL, CC low, n=0, 11, 0 |  | 0 |
  TNUE, TC 6, PBL, CC low, n=0, 11, 0 |  | 0 |
  TNUE, TC 6, BL, CC high, n=0, 11, 0 |  | 0 |
  TNUE, TC 6,PBL, CC high, n=0, 11, 0 |  | 0 |
  WBC count, TC 6, BL, CC low, n=0, 11, 0 |  | 0 |
  WBC count, TC 6, PBL, CC low, n=0, 11, 0 |  | 0 |
  WBC count, TC 6, BL, CC high, n=0, 11, 0 |  | 0 |
  WBC count, TC 6, PBL, CC high, n=0, 11, 0 |  | 0 |
  Eosinophils, TC 7, BL, CC high, n=0, 2, 0 |  | 0 |
  Eosinophils, TC 7, PBL, CC high, n=0, 2, 0 |  | 0 |
  HCT, TC 7, BL, CC low, n=0, 2, 0 |  | 0 |
  HCT, TC 7, PBL, CC low, n=0, 2, 0 |  | 0 |
  Hb, TC 7, BL, CC low, n=0, 2, 0 |  | 0 |
  Hb, TC 7, PBL, CC low, n=0, 2, 0 |  | 0 |
  Lymphocytes, TC 7, BL, CC low, n=0, 2, 0 |  | 0 |
  Lymphocytes, TC 7, PBL, CC low, n=0, 2, 0 |  | 0 |
  PC, TC 7, BL, CC high, n=0, 2, 0 |  | 0 |
  PC, TC 7, PBL, CC high, n=0, 2, 0 |  | 0 |
  RBC count, TC 7, BL, CC low, n=0, 2, 0 |  | 0 |
  RBC count, TC 7, PBL, CC low, n=0, 2, 0 |  | 0 |
  TNUE, TC 7, BL, CC low, n=0, 2, 0 |  | 0 |
  TNUE, TC 7, PBL, CC low, n=0, 2, 0 |  | 0 |
  TNUE, TC 7, BL, CC high, n=0, 2, 0 |  | 0 |
  TNUE, TC 7,PBL, CC high, n=0, 2, 0 |  | 0 |
  WBC count, TC 7, BL, CC low, n=0, 2, 0 |  | 0 |
  WBC count, TC 7, PBL, CC low, n=0, 2, 0 |  | 0 |
  WBC count, TC 7, BL, CC high, n=0, 2, 0 |  | 0 |
  WBC count, TC 7, PBL, CC high, n=0, 2, 0 |  | 0 |

43. Secondary Outcome: Number of Participants With the Indicated Biomarker Data Outside the Reference Range at Baseline or Any Post-Baseline Visit During the DB and OL Periods by Ofatumumab Treatment Course (TC)
Description: Only those parameters for a particular flag (<LLN or >ULN) are summarized if at least one value was outside the specified reference range. The Baseline (BL) value for a TC was defined as the latest value on or before the date of infusion A of the TC. However to be evaluable as a baseline value, assessments must have been conducted within a 14 day window prior to the date of infusion A. The post-baseline (PBL) was any visit after the date of infusion A during the specified TC. The pre-defined LLN for biomarkers are: B-lymphocyte stimulator (B-ls):<486.5 nanograms per Liter (ng/L); Interleukin-6 (IL-6):<0.31ng/L and Serum amyloid A: <1951 ng/mL. LLN was not defined for Rheumatoid factor (RF)-IgA, RF-IgG, RF-IgM or anti- cyclic citrullinated peptide (CCP) antibody and RF. The pre- defined ULN range for biomarkers (RF)-IgA: >6 units; RF-IgG:>6 units; RF-IgM:>6 units; Anti-CCP:>19.9999 units; B-ls:>1343.3 ng/L; IL-6: >5 ng/L; RF:>11.9999 kilounits (KU)/L; Serum amyloid A:>82432 ng/mL.
Time Frame: From baseline up to Week 144
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 205 | 0
Participants
  RF IgA, TC 1, BL, >ULN, n=0, 205, 0 |  | 137 |
  RF IgA, TC 1, PBL, >ULN, n=0, 169, 0 |  | 93 |
  RF IgG, TC 1, BL, >ULN, n=0, 205, 0 |  | 114 |
  RF IgG, TC 1, PBL, >ULN, n=0, 169, 0 |  | 67 |
  RF IgM, TC 1, BL, >ULN, n=0, 205, 0 |  | 173 |
  RF IgM, TC 1, PBL, >ULN, n=0, 169, 0 |  | 129 |
  Anti-CCP, TC 1, BL, >ULN, n=0, 207, 0 |  | 185 |
  Anti-CCP, TC 1, PBL, >ULN, n=0, 168, 0 |  | 140 |
  B-ls, TC 1, BL, <LLN, n=0, 203, 0 |  | 21 |
  B-ls, TC 1, PBL, <LLN, n=0, 206, 0 |  | 4 |
  B-ls, TC 1, BL, >ULN, n=0, 203, 0 |  | 12 |
  B-ls, TC 1, PBL, >ULN, n=0, 206, 0 |  | 167 |
  Il-6, TC 1, BL, >ULN, n=0, 205, 0 |  | 144 |
  IL-6, TC 1, PBL, >ULN, n=0, 138, 0 |  | 79 |
  Serum amyloid A, TC 1, BL, >ULN, n=0, 204, 0 |  | 129 |
  Serum amyloid A, TC 1, PBL, >ULN, n=0, 138, 0 |  | 68 |
  RF IgA, TC 2, BL, >ULN, n=0, 59, 0 |  | 32 |
  RF IgA, TC 2, PBL, >ULN, n=0, 111, 0 |  | 51 |
  RF IgG, TC 2, BL, >ULN, n=0, 59, 0 |  | 20 |
  RF IgG, TC 2, PBL, >ULN, n=0, 111, 0 |  | 38 |
  RF IgM, TC 2, BL, >ULN, n=0, 59, 0 |  | 45 |
  RF IgM, TC 2, PBL, >ULN, n=0, 111, 0 |  | 80 |
  Anti-CCP, TC 2, BL, >ULN, n=0, 60, 0 |  | 51 |
  Anti-CCP, TC 2, PBL, >ULN, n=0, 111, 0 |  | 93 |
  B-ls, TC 2, BL, <LLN, n=0, 81, 0 |  | 1 |
  B-ls, TC 2, PBL, <LLN, n=0, 88, 0 |  | 1 |
  B-ls, TC 2, BL, >ULN, n=0, 81, 0 |  | 60 |
  B-ls, TC 2, PBL, >ULN, n=0, 88, 0 |  | 72 |
  Il-6, TC 2, BL, >ULN, n=0, 52, 0 |  | 23 |
  IL-6, TC 2, PBL, >ULN, n=0, 23, 0 |  | 8 |
  Serum amyloid A, TC 2, BL, >ULN, n=0, 52, 0 |  | 18 |
  Serum amyloid A, TC 2, PBL, >ULN, n=0, 24, 0 |  | 4 |
  RF IgA, TC 3, BL, >ULN, n=0, 20, 0 |  | 9 |
  RF IgA, TC 3, PBL, >ULN, n=0, 95, 0 |  | 42 |
  RF IgG, TC 3, BL, >ULN, n=0, 20, 0 |  | 7 |
  RF IgG, TC 3, PBL, >ULN, n=0, 95, 0 |  | 21 |
  RF IgM, TC 3, BL, >ULN, n=0, 20, 0 |  | 14 |
  RF IgM, TC 3, PBL, >ULN, n=0, 95, 0 |  | 61 |
  Anti-CCP, TC 3, BL, >ULN, n=0, 20, 0 |  | 16 |
  Anti-CCP, TC 3, PBL, >ULN, n=0, 94, 0 |  | 78 |
  B-ls, TC 3, BL, <LLN, n=0, 16, 0 |  | 0 |
  B-ls, TC 3, PBL, <LLN, n=0, 4, 0 |  | 0 |
  B-ls, TC 3, BL, >ULN, n=0, 16, 0 |  | 14 |
  B-ls, TC 3, PBL, >ULN, n=0, 4, 0 |  | 4 |
  Il-6, TC 3, BL, >ULN, n=0, 0, 0 |  | 0 |
  IL-6, TC 3, PBL, >ULN, n=0, 21, 0 |  | 9 |
  Serum amyloid A, TC 3, BL, >ULN, n=0, 0, 0 |  | 0 |
  Serum amyloid A, TC 3, PBL, >ULN, n=0, 21, 0 |  | 4 |
  RF IgA, TC 4, BL, >ULN, n=0, 14, 0 |  | 6 |
  RF IgA, TC 4, PBL, >ULN, n=0, 43, 0 |  | 19 |
  RF IgG, TC 4, BL, >ULN, n=0, 14, 0 |  | 2 |
  RF IgG, TC 4, PBL, >ULN, n=0, 43, 0 |  | 13 |
  RF IgM, TC 4, BL, >ULN, n=0, 14, 0 |  | 8 |
  RF IgM, TC 4, PBL, >ULN, n=0, 43, 0 |  | 27 |
  Anti-CCP, TC 4, BL, >ULN, n=0, 14, 0 |  | 10 |
  Anti-CCP, TC 4, PBL, >ULN, n=0, 45, 0 |  | 35 |
  B-ls, TC 4, BL, <LLN, n=0, 0, 0 |  | 0 |
  B-ls, TC 4, PBL, <LLN, n=0, 0, 0 |  | 0 |
  B-ls, TC 4, BL, >ULN, n=0, 0, 0 |  | 0 |
  B-ls, TC 4, PBL, >ULN, n=0, 0, 0 |  | 0 |
  Il-6, TC 4, BL, >ULN, n=0, 0, 0 |  | 0 |
  IL-6, TC 4, PBL, >ULN, n=0, 18, 0 |  | 5 |
  Serum amyloid A, TC 4, BL, >ULN, n=0, 0, 0 |  | 0 |
  Serum amyloid A, TC 4, PBL, >ULN, n=0, 17, 0 |  | 4 |
  RF IgA, TC 5, BL, >ULN, n=0, 5, 0 |  | 1 |
  RF IgA, TC 5, PBL, >ULN, n=0, 24, 0 |  | 10 |
  RF IgG, TC 5, BL, >ULN, n=0, 5, 0 |  | 1 |
  RF IgG, TC 5, PBL, >ULN, n=0, 24, 0 |  | 5 |
  RF IgM, TC 5, BL, >ULN, n=0, 5, 0 |  | 4 |
  RF IgM, TC 5, PBL, >ULN, n=0, 24, 0 |  | 17 |
  Anti-CCP, TC 5, BL, >ULN, n=0, 5, 0 |  | 4 |
  Anti-CCP, TC 5, PBL, >ULN, n=0, 24, 0 |  | 20 |
  B-ls, TC 5, BL, <LLN, n=0, 0, 0 |  | 0 |
  B-ls, TC 5, PBL, <LLN, n=0, 0, 0 |  | 0 |
  B-ls, TC 5, BL, >ULN, n=0, 0, 0 |  | 0 |
  B-ls, TC 5, PBL, >ULN, n=0, 0, 0 |  | 0 |
  Il-6, TC 5, BL, >ULN, n=0, 0, 0 |  | 0 |
  IL-6, TC 5, PBL, >ULN, n=0, 5, 0 |  | 1 |
  Serum amyloid A, TC 5, BL, >ULN, n=0, 0, 0 |  | 0 |
  Serum amyloid A, TC 5, PBL, >ULN, n=0, 5, 0 |  | 1 |
  RF IgA, TC 6, BL, >ULN, n=0, 6, 0 |  | 0 |
  RF IgA, TC 6, PBL, >ULN, n=0, 9, 0 |  | 3 |
  RF IgG, TC 6, BL, >ULN, n=0, 6, 0 |  | 0 |
  RF IgG, TC 6, PBL, >ULN, n=0, 9, 0 |  | 1 |
  RF IgM, TC 6, BL, >ULN, n=0, 6, 0 |  | 3 |
  RF IgM, TC 6, PBL, >ULN, n=0, 9, 0 |  | 6 |
  Anti-CCP, TC 6, BL, >ULN, n=0, 6, 0 |  | 4 |
  Anti-CCP, TC 6, PBL, >ULN, n=0, 9, 0 |  | 8 |
  B-ls, TC 6, BL, <LLN, n=0, 0, 0 |  | 0 |
  B-ls, TC 6, PBL, <LLN, n=0, 0, 0 |  | 0 |
  B-ls, TC 6, BL, >ULN, n=0, 0, 0 |  | 0 |
  B-ls, TC 6, PBL, >ULN, n=0, 0, 0 |  | 0 |
  Il-6, TC 6, BL, >ULN, n=0, 0, 0 |  | 0 |
  IL-6, TC 6, PBL, >ULN, n=0, 2, 0 |  | 0 |
  Serum amyloid A, TC 6, BL, >ULN, n=0, 0, 0 |  | 0 |
  Serum amyloid A, TC 6, PBL, >ULN, n=0, 2, 0 |  | 0 |
  RF IgA, TC 7, BL, >ULN, n=0, 2, 0 |  | 2 |
  RF IgA, TC 7, PBL, >ULN, n=0, 0, 0 |  | 0 |
  RF IgG, TC 7, BL, >ULN, n=0, 2, 0 |  | 0 |
  RF IgG, TC 7, PBL, >ULN, n=0, 0, 0 |  | 0 |
  RF IgM, TC 7, BL, >ULN, n=0, 2, 0 |  | 1 |
  RF IgM, TC 7, PBL, >ULN, n=0, 0, 0 |  | 0 |
  Anti-CCP, TC 7, BL, >ULN, n=0, 2, 0 |  | 2 |
  Anti-CCP, TC 7, PBL, >ULN, n=0, 0, 0 |  | 0 |
  B-ls, TC 7, BL, <LLN, n=0, 0, 0 |  | 0 |
  B-ls, TC 7, PBL, <LLN, n=0, 0, 0 |  | 0 |
  B-ls, TC 7, BL, >ULN, n=0, 0, 0 |  | 0 |
  B-ls, TC 7, PBL, >ULN, n=0, 0, 0 |  | 0 |
  Il-6, TC 7, BL, >ULN, n=0, 0, 0 |  | 0 |
  IL-6, TC 7, PBL, >ULN, n=0, 0, 0 |  | 0 |
  Serum amyloid A, TC 7, BL, >ULN, n=0, 0, 0 |  | 0 |
  Serum amyloid A, TC 7, PBL, >ULN, n=0, 0, 0 |  | 0 |

44. Secondary Outcome: Number of Participants With Any Serious Adverse Event During the Follow-up Period
Description: A serious adverse event is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; or is a congenital anomaly/birth defect. Medical or scientific judgment should have been exercised in other situations. Refer to the general SAE module for a list of SAEs.
Time Frame: From the last scheduled visit in the DB or OL Period until B-cells and circulating IgG had returned to normal or baseline levels (or maximum of 2 years from Last Subject Last Visit [LSLV])
Population: Safety Follow-up Population: all participants who withdrew from the Double-blind Period and had evidence of contact with the site after the end of the Double-blind Period and all participants who withdrew or completed the Open-label Period and had evidence of contact with the site after their end of Open-label date.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 0 | 224
Participants |  |  | 13

45. Secondary Outcome: Number of Participants With Immunoglobulin Values Outside the Reference Range During the Follow-up Period
Description: The reference ranges for immunoglobulins (LLN, ULN) are defined as: IgA (grams/Liter): 0.81, 4.63; IgG (grams/Liter): 6.94, 16.18; IgM (grams/Liter): 0.48, 2.71.
Time Frame: From the last scheduled visit in the DB or OL Period until B-cells and circulating IgG had returned to normal or baseline levels (or maximum of 2 years from LSLV)
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 0 | 220
Participants
  IgA <LLN |  |  | 1
  IgA >ULN |  |  | 29
  IgG <LLN |  |  | 16
  IgG >ULN |  |  | 20
  IgM <LLN |  |  | 35
  IgM >ULN |  |  | 7

46. Secondary Outcome: Time to First CD19+ B-cell Repopulation Relative to the First Dose and Last Dose of Ofatumumab
Description: Time to first CD19+ B-cell repopulation (return to normal or baseline level) relative to the first dose was assessed only for those participants whose B-cells repopulated after receiving ofatumumab. Time to first CD19+ B-cell repopulation relative to the last dose of ofatumumab was assessed only for those participants whose B-cells repopulated during their last ofatumumab treatment course or follow-up.
Time Frame: From the first dose of ofatumumab until the last Follow-up Period visit (up to Week 248)
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Median (Full Range); unit: Months
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 0 | 133
Months
  Relative to first dose, n=0, 0, 133 |  |  | 22.998 [0.43 to 56.64]
  Relative to last dose, n=0, 0, 128 |  |  | 13.832 [3.06 to 54.77]

47. Secondary Outcome: Number of Participants With a Positive JC Virus Test Result During the Follow-up Period
Description: Blood samples were collected for analysis of plasma/white blood cell JC Virus (JCV) using the polymerase chain reaction (PCR) assay. A positive JC Virus test result indicated the presence of JC Virus.
Time Frame: as for outcome 45
Population: AT Population. Only those participants contributing values at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 0 | 243
Participants |  |  | 8

48. Secondary Outcome: Number of Participants With the Indicated Clinical Chemistry Values of Potential Clinical Concern During the Follow-up Period
Description: Only those parameters for which at least one value of clinical concern (CC) was reported are summarized. Pre-defined limits of potential clinical concern (CC Low [relative to the lower limit of normal], CC High [relative to the upper limit of normal]) are: ALT: NA, 2; ALP: NA, 1.5; Creatinine: N/A, 1.2; CO2/BCO: 0.85/0.75, 1.2/1.3; CK: NA, 2; GGT: NA, 2; Urea/BUN: NA, 1.5.
Time Frame: From the last scheduled visit in the DB or OL Period until B-cells and circulating IgG had returned to normal or baseline levels (maximum of 2 years)
Population: AT Population. Only participants who withdrew from the DB Period and had evidence of contact with the site after the end of the DB Period and all participants who withdrew or completed the OL Period and had evidence of contact with the site after their end of OL date were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 0 | 224
Participants
  ALT |  |  | 1
  ALP |  |  | 1
  CK |  |  | 2
  CO2/BCO |  |  | 3
  GGT |  |  | 5
  Creatinine |  |  | 1
  Urea/BUN |  |  | 1

49. Secondary Outcome: Number of Participants With the Indicated Hematology Values of Potential Clinical Concern During the Follow-up Period
Description: Only those parameters for which at least one value of clinical concern (CC) was reported are summarized. Pre-defined limits of potential clinical concern (CC Low [relative to lower limit of normal], CC High [relative to upper limit of normal]) are: Eosinophils: NA, 2; Total neutrophils: 0.8, 1.6; Platelet count: 0.65, 1.5.
Time Frame: as for outcome 48
Population: as for outcome 48
Measure: Number; unit: Participants
Arm/Group | Placebo | Ofatumumab 700 mg | Placebo or OFA 700 mg: FU Period
Number analyzed (Participants) | 0 | 0 | 224
Participants
  Eosinophils |  |  | 1
  Total neutrophils |  |  | 2
  Platelet count |  |  | 1

ADVERSE EVENTS:
Time Frame: Because no investigational product was administered during the Follow-up Period, per protocol, only serious adverse events (SAEs) were collected and reported for this period.
Description: SAEs/AEs were collected in members of the Safety Population (SP), which is identical to the ITT Population, except that participants were analyzed according to the actual treatment received rather than to the treatment randomized to (one participant was randomized to placebo but received study drug).
Groups:
- Placebo: DB Period: Serious adverse events (SAEs) and non-serious AEs are reported for participants receiving placebo in the DB Period. Placebo was administered as two 1000 milliliter (ml) intravenous (IV) infusions, one at Day 0 and the other at Day 14, in addition to background methotrexate (MTX) treatment (7.5 to 25 milligrams [mg]/week [oral, intramuscular, or subcutaneous] for 24 weeks) in the DB Period.
- Ofatumumab 700 mg: DB and OL Periods: SAEs and non-serious AEs are reported for participants receiving ofatumumab 700 mg in either the DB or OL Period. Ofatumumab 700 mg (35 ml) was administered as two 1000 ml IV infusions, one at Day 0 and the other at Day 14, in addition to background MTX treatment (7.5 to 25 mg/week [oral, intramuscular, or subcutaneous] for 24 weeks) in the DB Period. Participants completing the 24-week DB Period without receiving rescue disease-modifying anti-rheumatic drug treatment were eligible to proceed into the 120-week OL Period to receive repeat ofatumumab treatment courses (at individualized time intervals if a clinical response had been achieved after the previous treatment course).
- Placebo or Ofatumumab 700 mg: Follow-up Period: SAEs and non-serious AEs are reported for participants receiving either placebo or ofatumumab 700 mg in the Follow-up Period. Participants randomized to DB treatment who completed the OL Period, who did not enter the OL Period, who did not qualify for retreatment, or who were withdrawn were to be followed until the number of B-cells and circulating IgG had returned to normal (according to the central laboratory) or Baseline levels or for a maximum of 2 years from the last scheduled visit in the DB or OL Periods, whichever occurred earlier. No investigational product was administered in the Follow-up Period.
Arm/Group | Placebo: DB Period | Ofatumumab 700 mg: DB and OL Periods | Placebo or Ofatumumab 700 mg: Follow-up Period
Serious Adverse Events (participants affected / at risk) | 4/130 | 44/243 | 13/224
Other Adverse Events (participants affected / at risk) | 46/130 | 226/243 | 0/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: DB Period (N=130) | Ofatumumab 700 mg: DB and OL Periods (N=243) | Placebo or Ofatumumab 700 mg: Follow-up Period (N=224)
Pneumonia (Infections and infestations) | 1 | 1 | 0
Gastroenteritis bacterial (Infections and infestations) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 2 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Axillary vein thrombosis (Vascular disorders) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Blepharospasm (Eye disorders) | 0 | 1 | 0
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cardiac aneurysm (Cardiac disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1 | 0
Colonic stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0
Endometritis (Infections and infestations) | 0 | 1 | 0
Gingival cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pertusis (Infections and infestations) | 0 | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0
Post cholecystectomy syndrome (Hepatobiliary disorders) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Troponin T increased (Investigations) | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pancreatic necrosis (Gastrointestinal disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: DB Period (N=130) | Ofatumumab 700 mg: DB and OL Periods (N=243) | Placebo or Ofatumumab 700 mg: Follow-up Period (N=224)
Rash (Skin and subcutaneous tissue disorders) | 1 | 89 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 45 | 0
Urinary tract infection (Infections and infestations) | 9 | 27 | 0
Headache (Nervous system disorders) | 8 | 20 | 0
Nasopharyngitis (Infections and infestations) | 3 | 34 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 26 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 43 | 0
Hypertension (Vascular disorders) | 5 | 20 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 15 | 0
Hypersensitivity (Immune system disorders) | 0 | 11 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 20 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 9 | 0
Anaemia (Blood and lymphatic system disorders) | 5 | 9 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 20 | 0
Nausea (Gastrointestinal disorders) | 4 | 13 | 0
Bacteriuria (Infections and infestations) | 2 | 5 | 0
Influenza (Infections and infestations) | 4 | 8 | 0
Leukocyturia (Renal and urinary disorders) | 2 | 9 | 0
Pharyngitis (Infections and infestations) | 1 | 13 | 0
Bronchitis (Infections and infestations) | 4 | 18 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 24 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 5 | 0
Haematuria (Renal and urinary disorders) | 1 | 10 | 0
Alanine aminotransferase increased (Investigations) | 4 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 12 | 0
Dizziness (Nervous system disorders) | 1 | 7 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 13 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 | 7 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 9 | 0
Gastroenteritis (Infections and infestations) | 0 | 9 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 9 | 0
Depression (Psychiatric disorders) | 0 | 8 | 0
Gastritis (Gastrointestinal disorders) | 0 | 8 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 8 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 8 | 0
Sinusitis (Infections and infestations) | 0 | 7 | 0
Blood pressure increased (Investigations) | 0 | 6 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 6 | 0
Cellulitis (Infections and infestations) | 0 | 6 | 0
Conjunctiviitis (Eye disorders) | 0 | 6 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 6 | 0
Flushing (Vascular disorders) | 0 | 6 | 0
Lymphocyte count decreased (Investigations) | 0 | 6 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 6 | 0
Oedema peripheral (General disorders) | 0 | 6 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0
Tachycardia (Cardiac disorders) | 0 | 6 | 0
Vomiting (Gastrointestinal disorders) | 0 | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0
Chest pain (General disorders) | 0 | 5 | 0
Drug intolerance (General disorders) | 0 | 5 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 5 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 5 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 5 | 0
Sciatica (Nervous system disorders) | 0 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.